# A Prospective, Multi-center and Noninferiority Clinical Study Evaluating Trochanteric Fixation Nail Advanced (TFNA) in Chinese Patient Population

# Statistical Analysis Plan

# V1.3

Statistical institution: Medical Research & Biometrics Center, National

**Center for Cardiovascular Diseases** 

Sponsor: Johnson & Johnson Medical (Shanghai) Ltd.

Date of issue: May 19, 2020

## **Confidential Statement**

The information contained in this document is proprietary and confidential. Any reproduction, dissemination or distribution, in whatever form and by whatever media, is expressly prohibited without the prior written consent of the contact person of Johnson & Johnson Medical (Shanghai) Ltd.

# **Signature Page**

| Study title: | A Prospective, Multi-center and Non-inferiority Clinical Study Evaluating<br>Trochanteric Fixation Nail Advanced (TFNA) in Chinese Patient Population | |
|---|---|---|
| Sponsor: | Johnson & Johnson Medical (Shanghai) Co., Ltd. | |
| Study No.: | DPS-201502 | |
| Date of issue: | May 19, 2020 | |
| Version No.: | V1.3 | |
| Sponsor/CRO | Title: | MM/DD/YYYY |
| Principal investigator (PI) | Title: | MM/DD/YYYY |
| Author of the Plan (NCCD) | Title: | MM/DD/YYYY |
| Plan review (NCCD) | Title: | MM/DD/YYYY |

# **Table of Contents**

| Ch | apte | er | Page |
|---|---|---|---|
| Sign | nature | e Page | 1 |
| | | obreviations and Definitions of Terms | |
| 1. | Intro | oduction | 7 |
| 2. | Clini | cal Study | 7 |
| | 2.1 | Study objective | 7 |
| | 2.2 | Study design | 7 |
| | 2.3 | Primary endpoint | 8 |
| | 2.4 | Secondary endpoints | |
| <b>3.</b> | Inves | stigational Device | |
| | 3.1 | Investigational device | |
| | 3.2 | Control device | |
| 4. | | ded Use and Indications of the Product | |
| 5. | Inclu | sion and Exclusion Criteria of Subjects | |
| | 5.1 | Inclusion criteria | |
| | 5.2 | Exclusion criteria | |
| 6. | | eral Statistical Considerations | |
| | 6.1 | Study hypothesis | |
| | 6.2 | Sample size calculation | |
| | 6.3 | Analysis population | |
| | 6.4 | Detailed rules for determination of analysis population set and flow chart | |
| | 6.5 | Missing values, abnormal values and outlying values | |
| | 6.6 | Significant level and statistical analysis software | |
| _ | 6.7 | Site merging principle | |
| 7. | | stical Analysis Indicators and Statistical Analysis Methods | 16 |
| | 7.1 | Demographic indicators and other baseline indicators | |
| | 7.2 | Intraoperative information | |
| | 7.3 | Primary endpoint | |
| | 7.4 | Secondary endpoints | |
| | 7.5 | Follow-up data | |
| | 7.6<br>7.7 | Laboratory examinations | |
| 0 | | Concomitant medication, adverse events (AEs) or serious adverse events (SAEs) | |
| 8.<br>Fig. | Gene<br>ure 1 | Flow chart for determination of analysis population data sets | |
| Tab | | Determination of analysis population | 25<br>26 |
| | ole 1 | List of subjects who withdrawal the informed consent or seriously violate the | |
| | 27 | List of subjects who withdrawar the informed consent of seriously violate the | protocor |
| Tab | | List of subjects who violate the protocol (CRF collection) | 28 |
| Tab | | Determination of analysis population in Beijing Jishuitan Hospital | |
| | le 5 | Determination of analysis population in Peking University Third Hospital | |
| | le 6 | Determination of analysis population in Chinese PLA General Hospital | |
| Tab | | Determination of analysis population in the Second Affiliated Hospital of Z | |
| | | y School of Medicine | |
| | le 8 | Determination of analysis population in Shanghai General Hospital | |
| | le 9 | Determination of analysis population in Nanfang Hospital Of Southern | |
| | versit | • • • | 1110411041 |
| | le 10 | Determination of analysis population in Affiliated Hospital of Nantong University | sity35 |
| | le 11 | Determination of analysis population in West China Hospital, Sichuan Univers | • |
| | le 12 | Determination of analysis population in the First Affiliated Hospital of Gu | |
| | | y of Chinese Medicine | _ |
| | le 13 | Determination of analysis population in the University of Hong Kong - S | |
| | pital | 38 | |
| | le 14 | Statistical analysis results of subjects' demographic data | 39 |

| Table 15 | Statistical analysis results of subjects' height and body weight4 | 0 |
|---|---|---|
| Table 16 | Statistical analysis results of subjects' previous and current medical history4 | 1 |
| Table 16 | Statistical analysis results of subjects' previous and current medical history (continue | d |
| 1) 43 | | |
| Table 16 | Statistical analysis results of subjects' previous and current medical history (continue | d |
| 2) 44 | | |
| Table 17 | Statistical analysis results of subjects' preoperative SF-12v2 questionnaire4 | 5 |
| Table 17 | Statistical analysis results of subjects' preoperative SF-12v2 questionnaire (continued | l) |
| 46 | | |
| Table 18 | Statistical analysis results of subjects' preoperative EQ-5D questionnaire4 | 7 |
| Table 18 | Statistical analysis results of subjects' preoperative EQ-5D questionnaire (continued | I) |
| 48 | | |
| Table 19 | Statistical analysis results of subjects' preoperative fractures4 | 9 |
| Table 20 | Statistical analysis results of subjects' x-ray examination before surgery5 | 0 |
| Table 21 | Statistical analysis results of subjects' use of investigational devices5 | 1 |
| Table 21 | Statistical analysis results of subjects' use of investigational devices (continued)5 | 2 |
| Table 22 | Statistical analysis results of subjects' use of other devices5 | 3 |
| Table 23 | Statistical analysis results of subjects' surgical details5 | 4 |
| Table 24 | Statistical analysis results of subjects' intraoperative fractures5 | 5 |
| Table 24 | Statistical analysis results of subjects' intraoperative fractures (continued)5 | 6 |
| Table 25 | Statistical analysis results of subjects' evaluation on product operability and tool | S |
| during the su | ırgery5 | |
| Table 26 | Statistical analysis results of subjects' intraoperative AEs5 | |
| Table 27 | Statistical analysis results of subjects' intraoperative medication records5 | |
| Table 28 | Statistical analysis results of subjects' intraoperative combination therapy6 | |
| Table 29 | (FAS) Primary endpoint - statistical analysis results of fracture union rate of subjects a | ıt |
| | veeks after surgery6 | |
| Table 29 | (FAS) Primary endpoint - statistical analysis results of fracture union rate of subjects a | |
| | veeks after surgery (continued)6 | |
| Table 30 | (FAS) Primary endpoint - Statistical analysis results of subjects' fracture union rate 2 | |
| | urgery6 | |
| Table 31 | (PPS) Primary endpoint - statistical analysis results of fracture union rate of subjects a | |
| | weeks after surgery6 | |
| Table 31 | (PPS) Primary endpoint - statistical analysis results of fracture union rate of subjects a | |
| | weeks after surgery (continued)6 | |
| Table 32 | (PPS) Primary endpoint - Statistical analysis results of subjects' fracture union rate 2 | |
| | urgery6 | 6 |
| Table 33 | (ATS) Primary endpoint - Statistical analysis results of subjects' fracture union rate 2 | |
| | urgery6 | |
| Table 34 | (FAS) Secondary endpoint - Statistical analysis results of adverse events of subjects 6 | |
| Table 35 | (FAS) Secondary endpoint - Statistical analysis results of subjects' revision rate 2 | |
| | urgery6 | |
| Table 36 | (FAS) Secondary endpoint - Statistical analysis results of subjects' re-operation rate 2 | |
| | urgery | |
| Table 37 | (FAS) Secondary endpoint - Statistical analysis results of subjects' Harris hip score 1 | |
| | urgery | 1 |
| Table 38 | (FAS) Secondary endpoint - Statistical analysis results of subjects' Harris hip score 2 | |
| Table 39 | urgery | |
| Table 39 | e 12 weeks after surgery | |
| | e 12 weeks after surgery (continued 1) | |
| Table 39 | (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v | |
| | e 12 weeks after surgery (continued 2) | |
| Table 39 | (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v | |
| | e 12 weeks after surgery (continued 3) | |
| _ | urch & Biometrics Center, National Version No.: V1.0 3/129 | |
| | J/12) | |

| Table 40 | (FAS) Secondary endpoint - Statistic | | |
|---|---|---|---|
| questionnaire | e 24 weeks after surgery | •••••• | 79 |
| Table 40 | (FAS) Secondary endpoint - Statistic | cal analysis results of subjects | ' SF-12v2 |
| questionnaire | e 24 weeks after surgery (continued 1) | | 80 |
| Table 40 | (FAS) Secondary endpoint - Statistic | cal analysis results of subjects | ' SF-12v2 |
| questionnaire | e 24 weeks after surgery (continued 2) | - | 82 |
| Table 40 | (FAS) Secondary endpoint - Statistic | cal analysis results of subjects | ' SF-12v2 |
| questionnaire | e 24 weeks after surgery (continued 3) | | |
| Table 41 | (FAS) Secondary endpoint - Statistical and | alysis results of subjects' EQ-5D que | estionnaire |
| 12 weeks afte | er surgery | | |
| Table 41 | (FAS) Secondary endpoint - Statistical and | alysis results of subjects' EQ-5D qu | estionnaire |
| | er surgery(continue) | | |
| Table 42 | (FAS) Secondary endpoint - Statistical and | alysis results of subjects' EO-5D que | estionnaire |
| | er surgery | | 87 |
| Table 42 | (FAS) Secondary endpoint - Statistical an | alysis results of subjects' EO-5D que | estionnaire |
| | er surgery(continue) | | |
| Table 43 | (FAS) Secondary endpoint - Statistical a | | |
| | s requiring re-operation or revision | · · | |
| Table 44 | (PPS) Secondary endpoint - Statistical an | alysis results of subjects' AE | 90 |
| Table 45 | (PPS) Secondary endpoint - Statistical and | | |
| after surgery | | ay sistes are subjects for island | te 21 weeks |
| Table 46 | (PPS) Secondary endpoint - Statistical an | alvsis results of subjects' re-onerat | ion rate 24 |
| | surgery | | |
| Table 47 | (PPS) Secondary endpoint - Statistical ar | alvsis results of subjects, Harris b | |
| | Surgery | | |
| Table 48 | (PPS) Secondary endpoint - Statistical ar | alveie results of subjects? Harris b | |
| | • • | · · | - |
| | surgery(FAS) Secondary endpoint - Statistic | | |
| Table 49 | ` ' | · · | |
| - | e 12 weeks after surgery(PPS) Secondary endpoint - Statistic | | |
| Table 49 | | | |
| - | e 12 weeks after surgery (continued 1)<br>(PPS) Secondary endpoint - Statistic | | |
| Table 49 | • • | · | |
| - | te 12 weeks after surgery (continued 2) | | |
| Table 49 | (PPS) Secondary endpoint - Statistic | | |
| - | e 12 weeks after surgery (continued 3) | | |
| Table 50 | (PPS) Secondary endpoint - Statistic | | |
| - | e 24 weeks after surgery | | 101 |
| Table 50 | (PPS) Secondary endpoint - Statistic | | |
| - | e 24 weeks after surgery (continued 1) | 1 1 . 1 | 102 |
| Table 50 | (PPS) Secondary endpoint - Statistic | | |
| • | e 24 weeks after surgery (continued 2) | | |
| Table 50 | (PPS) Secondary endpoint - Statistic | | |
| | e 24 weeks after surgery (continued 3) | | |
| Table 51 | (PPS) Secondary endpoint - Statistical and | | |
| | er surgery | | |
| Table 51 | (PPS) Secondary endpoint - Statistical and | | |
| | er surgery(continue) | | |
| Table 52 | (PPS) Secondary endpoint - Statistical and | | |
| | er surgery | | |
| Table 52 | (PPS) Secondary endpoint - Statistical and | | |
| | er surgery(continue) | | |
| Table 53 | (PPS) Secondary endpoint - Statistical a | | |
| | s requiring re-operation or revision | | |
| Table 54 | Statistical analysis results of subjects' AE | | |
| Table 55 | Statistical analysis results of subjects' me | | |
| Table 56 | Statistical analysis results of subjects' cor | nbination therapy 1 week after surg | gery114 |
| Medical Resea | arch & Biometrics Center, National | Version No.: V1.0 | 4/129 |

| Table 57 | Statistical analysis results of subjects' fractures 1 week after surgery | 115 |
|---|---|---|
| Table 58 | Statistical analysis results of subjects' x-ray examination at the fracture site | 1 week after |
| surgery | 116 | |
| Table 59 | Statistical analysis results of subjects' AE evaluation 6 weeks after surgery. | 117 |
| Table 60 | Statistical analysis results of subjects' medication records 6 weeks after sur | |
| Table 61 | Statistical analysis results of subjects' combination therapy 6 weeks after su | |
| Table 62 | Statistical analysis results of subjects' fractures 6 weeks after surgery | |
| Table 63 | Statistical analysis results of subjects' X-ray examination at the fracture | |
| after surgery | · | , |
| Table 64 | Statistical analysis results of subjects' AE evaluation 12 weeks after surgery | <b>122</b> |
| Table 65 | Statistical analysis results of subjects' medication records 12 weeks after su | |
| Table 66 | Statistical analysis results of subjects' combination therapy 12 weeks after s | |
| Table 67 | Statistical analysis results of subjects' fractures 12 weeks after surgery | |
| Table 68 | Statistical analysis results of subjects' X-ray examination at the fracture si | |
| after surgery | | ite 12 weeks |
| Table 69 | Statistical analysis results of subjects' AE evaluation 24 weeks after surgery | , 127 |
| Table 70 | Statistical analysis results of subjects' Me evaluation 24 weeks after su Statistical analysis results of subjects' medication records 24 weeks after su | |
| Table 70 | Statistical analysis results of subjects' medication records 24 weeks after su<br>Statistical analysis results of subjects' combination therapy 24 weeks after su | 0 1 |
| Table 71 | Statistical analysis results of subjects' combination therapy 24 weeks after surgery | 0 . |
| Table 72 | | |
| | Statistical analysis results of subjects' x-ray examination at the fracture si | ite 24 weeks |
| after surgery | | hafana and |
| Table 74 | Statistical analysis results of outcomes of subjects' complete blood count | |
| | (before surgery → immediately after surgery) | |
| Table 74 | Statistical analysis results of outcomes of subjects' complete blood count | |
| | (before surgery → immediately after surgery) (continued) | |
| Table 75 | List of subjects with abnormal complete blood count with clinical signifi | |
| surgery chan<br>136 | ged from normal indicators before surgery (before surgery $ ightarrow$ immediately af | ter surgery) |
| Table 76 | Statistical analysis results of outcomes of subjects' blood biochemical test | before and |
| after surgery | (before surgery → immediately after surgery) | 137 |
| Table 76 | Statistical analysis results of outcomes of subjects' blood biochemical test | before and |
| after surgery | (before surgery $\rightarrow$ immediately after surgery) (continued 1) | 139 |
| Table 76 | Statistical analysis results of outcomes of subjects' blood biochemical test | before and |
| after surgery | (before surgery $\rightarrow$ immediately after surgery) (continued 2) | 141 |
| Table 77 | List of subjects with abnormal blood biochemical test indicators w | ith clinical |
| significance | after surgery changed from normal indicators before surgery (before | |
| | after surgery) | |
| Table 78 | List of concomitant medication of subjects | |
| Table 79 | Specific description on subjects with AEs | |
| Table 80 | Summary of AEs. | |
| Table 80 | Summary of AEs (continued 1) | |
| Table 81 | Specific description on subjects with investigational device-related AEs | |
| Table 82 | Summary of investigational device-related AEs | |
| Table 82 | Summary of investigational device-related AEs (continued) | |
| Table 83 | Summary of AEs (Number of events per subject) | |
| Table 84 | Statistical analysis results of the severity and the device related AEs (Accord | |
| 151 | Statistical analysis results of the severity and the device related ALS (Accord | ing subject) |
| Table 85 | Statistical analysis results of the severity and the device related AEs (Numb | er of events |
| per subject) | 152 | ci di events |
| Table 86 | Specific description on subjects with SAEs | 154 |
| Table 87 | Summary of SAEs | |
| Table 87 | Summary of SAEs (continued) | |
| Table 88 | Specific description on subjects with investigational device-related SAEs | |
| Table 89 | Summary of investigational device-related SAEs | |
| Table 89 | Summary of investigational device-related SAEs (continued) | |
| | Summary of investigational device-related SAEs (continued) | |
| Table 90 | • | |
| Medical Resea | rch & Biometrics Center, National Version No.: V1.0 | 5/129 |

| Table 91 | Statistical analysis results of the severity and the device related SAEs (Aco | cording subject) |
|---|---|---|
| 161 | | , |
| Table 92 | Statistical analysis results of the severity and the device related SAEs (No | umber of events |
| per subject) | 162 | |
| Table 93 | Specific description on subjects with UADEs | 164 |
| Table 94 | Summary of UADEs | 165 |
| Table 94 | Summary of UADEs (continued) | 166 |

## List of Abbreviations and Definitions of Terms

| Abbreviation | Definition |
|---|---|
| GCP | Good Clinical Practice |
| CRF | Case Report Form |
| SF-12 | 12-Item Short Form Health Survey |
| IRB | Institutional Review Board |
| EC | <b>Ethics Committee</b> |
| ERB | Ethical Review Board |
| BMI | <b>Body Mass Index</b> |
| AE | Adverse Event |
| SAE | Serious Adverse Event |
| <b>UADE</b> | <b>Unanticipated Adverse Device Effect</b> |
| ICH-GCP | International Conference on<br>Harmonization - Good Clinical Practice |
| HHS | Harris Hip Score |
| EQ5D | EuroQol-5D |

### 1. Introduction

This document provides the specific contents of the statistical analysis plan for a prospective, multi-center and non-inferiority clinical study on the safety and effectiveness of Trochanteric Fixation Nail Advanced (TFNA) manufactured by Johnson & Johnson Medical (Shanghai) Ltd. After all subjects are included and use the implant, the postoperative 24-week (±4 weeks) follow-up is completed or the trial is terminated in advance and the database is forcibly locked, the statistical analysis report for preoperative preparation and postoperative 24-week (±4 weeks) follow-up will be issued for registration application. Refer to the relevant tables, lists and graphs in the statistical analysis plan for the detailed specific analysis.

## 2. Clinical Study

## 2.1 Study objective

The primary objective of this study is to evaluate whether fracture union rate, evaluated 24 weeks after proximal femur fracture, for the investigational TFNA intramedullary nail is non-inferior to that for currently available control product PFNA-II in patients with proximal femur fractures.

## 2.2 Study design

The Trochanteric Fixation Nail Advanced (TFNA) is an implant designed to treat

proximal femur fractures and is currently in use in several regions worldwide (e.g., US, Europe). TFNA is manufactured using a titanium-molybdenum alloy (TiMo) that has not been used for a similar clinical application within China. The study is a prospective, multi-center, controlled, two-arm, randomized, non-inferiority study comparing the 24-week fracture union rate for proximal femur fractures treated with intramedullary nails using investigational devices (TFNA) compared to control devices (Proximal Femoral Nail Antirotation, PFNA-II), under a 10% non-inferiority margin.

## 2.3 Primary endpoint

The primary endpoint is the fracture union rate 24 weeks after surgery. Fracture union success is a composite endpoint; in order for an individual subject's surgery implanted with TFNA or PFNA-II to be considered successful he/she must satisfy all of the following criteria:

- 1. No focal tenderness or lengthwise percussion pain, or abnormal movement
- 2. The frontal/lateral X-ray examination shows the vague or no fracture gap, or the continuous callus passing across the fracture line
- 3. No deformation or breakage is found in the investigational product

## 2.4 Secondary endpoints

Secondary endpoints include the safety and effectiveness results, imaging outcomes and adverse events.

- Adverse events (type and frequency) for all adverse events will be compared for the study and control groups
- 24-week revision rate where revision is defined as removal of any component for any reason
- 24-week reoperation rate is defined as secondary surgery at the fracture site(s) for any reason
- Clinical Outcomes
- > SF-12
- ➤ Harris Hip Score
- ➤ EQ-5D
- Radiographs: incidence of complications such as loosening or cut-out that require reoperation or revision.

# 3. Investigational Device

# 3.1 Investigational device

- ➤ Short nails available in various diameters (Ø9, Ø10, Ø 11, Ø12 mm), lengths (170, 200, or 235 mm) and CCD angle (125°, 130° and 135°). The 235 mm short nail is available for left and right sides.
- Long nails available in various diameters (Ø9, Ø10, Ø 11, Ø12, Ø14mm), lengths (260-480mm in 20mm increments) and CCD angle (125°, 130° and 135°). All long nails are available for left and right sides.
- ➤ Head elements are available in blade and screw (both are 70-130 mm in length, available in 5mm increments)
- Locking screws (4.2mm diameter and available in lengths from 26-80mm (2mm increments) or 80-100mm (5mm increments)
- End caps available in 0, 5, 10 and 15mm lengths

## 3.2 Control device

PFNA-II as control product for this study, including:

- ➤ Short nails available in various diameters (Ø9, Ø10, Ø 11, Ø12 mm), lengths (170, 200, or 240 mm) and CCD angle (125° and 130°). The 240 mm short nail is available for left and right sides.
- ➤ Long nails available in various diameters (Ø9 and Ø10mm), lengths (260-340mm in 20mm increments and 340-420mm in 40mm increments) and CCD angle (125° and 130°). All long nails are available for left and right sides.
- ➤ Head elements are available in blade (70-120 mm in length, available in 5mm increments)
- Locking screws (4mm diameter and available in lengths from 16-60mm (2mm increments), 60-80mm (4mm increments) or 80-100mm (5mm increments)
- End caps available in 0, 5, 10 and 15mm lengths

## 4. Intended Use and Indications of the Product

## The intended use for TFNA is the following:

Intended Use: intended for the treatment of proximal femur and combinations of proximal and shaft fractures of the femur

## The indications of the TFNA are:

- Short Nails (lengths 170 mm, 200 mm, 235 mm)
- Pertrochanteric fractures (31-A1 and 31-A2)
- Intertrochanteric fractures (31-A3)
- 235 mm nails are additionally indicated for high subtrochanteric fractures

- Long Nails (lengths 260 mm 480 mm)
- Pertrochanteric fractures (31-A1 and 31-A2)
- Intertrochanteric fractures (31-A3)
- Fractures of the trochanteric area (31-A1/A2/A3) with diaphyseal extension
- Combined fractures of the trochanteric area (31-A1/A2/A3) and the femoral shaft (32-A/B/C)
- Pathological fractures, including prophylactic use
- Malunion
- Nonunion

## 5. Inclusion and Exclusion Criteria of Subjects

## 5.1 Inclusion criteria

# Subjects who meet all of the following inclusion criteria will be eligible for participation in the study:

- 1) Age  $\geq$ 18 years
- 2) Patients with unilateral proximal femur fractures that will be treated with intramedullary nail internal fixation
- 3) According to AO fracture classification, subjects with following fracture type:
- a. Pertrochanteric (31-A1 and 31-A2)
- b. Intertrochanteric (31-A3)
- c. Trochanteric area (31-A1/A2/A3) with diaphyseal extension
- 4) Subject must be comfortable with speaking and understanding questions and responses in an available translated language for patient reported outcomes (PROs)

### 5.2 Exclusion criteria

# Subjects who meet any of the following criteria will be excluded from the study:

- 1) Subject does not provide voluntary consent to participate in the study.
- 2) The subject is a woman who is pregnant or lactating
- 3) Fractures where the operative treatment will occur more than three weeks after the primary injury
- 4) Patients with femoral head fractures and femoral neck fractures (AO classification 31-B and 31-C)

- 5) Pathological fracture (e.g., primary or metastatic tumor)
- 6) Serious soft tissue injury, judged by the investigator, will impact the union of the fracture, combined vascular injury, and combined osteofascial compartment syndrome.
- 7) Multiple systemic injuries judged by researchers not suitable for enrollment, or orthopaedic fractures in other bones at three or more sites
- 8) Revision surgeries (for example, due to malunion, nonunion or infection)
- 9) Concurrent medical conditions judged by researchers not suitable for enrollment, such as: diabetes, metabolic bone disease, post-polio syndrome, poor bone quality, prior history of poor fracture healing, etc.
- 10) Patients with anaesthetic and surgical contraindications
- 11) Patents known to be allergic to implant components
- 12) Patients who are currently using chemotherapeutics or accepting radiotherapy, use systematically corticosteroid hormone or growth factor, or long-term use sedative hypnotics (continuous use over 3 months) or non-steroidal anti-inflammatory drugs (continuous use over 3 months)
- 13) Intemperance judged by researchers not suitable for enrollment (e.g., excessive daily drinking or smoking, drug abuse);
- 14) Patients participated into other clinical trial in the previous 3 months;
- 15) Patients with bad compliance judged by researchers and cannot complete the trial according to the study plan, such as schizophrenia and dementia.

## 6. General Statistical Considerations

## 6.1 Study hypothesis

The primary endpoint analysis will be to demonstrate that the investigational device (TFNA) is non-inferior to the control device (PFNA-II) based on the fracture union rates at the 24 week follow-up visit. Non-inferiority test will be conducted based on a one-sided 97.5% confidence interval for the difference in the fracture union rate at 24 weeks between the study group and the control group.

The primary hypothesis is that, at 24 weeks after surgery, the investigational device (TFNA) is non-inferior to the control device (PFNA-II) based on the individual patient fracture union rate. Non-inferiority is defined by a test with a two sided 5% type I error and a 10% "margin of non-inferiority".

Version No.: V1.0

The study's null and alternative hypotheses are as follows:

$$H_o: P_{PFNA-II} - P_{TFNA} \ge 10\%$$
  
 $H_a: P_{PFNA-II} - P_{TFNA} < 10\%$ 

Where, P<sub>PFNA-II</sub> represents the fracture union rate among those receiving PFNA-II implant and P<sub>TFNA</sub> denotes the fracture union rate among the recipients of TFNA.

Decision Criterion: The decision will be made to reject the null hypothesis  $H_0$  and conclude the alternative hypothesis  $H_a$  if the one-sided 97.5% confidence interval for the difference in the fracture union rates between the control group and the study group is less than the margin of non-inferiority, 10%.

## 6.2 Sample size calculation

The sample size calculation is determined based on the primary endpoint using PROC POWER in SAS software version 9.3. It assumes that the fracture union rate at 24 weeks after surgery in the TFNA group would be equivalent to that of the PFNA-II group, and a common fracture union rate is approximately 95% or greater based on the literature review. With a non-inferiority margin of 0.10 and a power of 80%, this implies a sample size of 75 for the TFNA and of 75 for PFNA-II surgery groups, respectively. The sample size will be increased to 188 (94 per group) to accommodate potential 20% attrition.

The sample size applies to patients enrolled, randomized, and actually treated. Some patients who enroll in a study and are randomized may not be ultimately treated for various reasons. Patient enrollment and randomization will continue until the proposed sample size for treated patients is complete.

## 6.3 Analysis population

Full Analysis Set (FAS): The set of subjects determined following the intent-totreat (ITT) principle refers to the data set constituted by all subjects who participate in the randomized study and receive the investigational product (implant) (i.e., ITT population defined in the protocol).

Per Protocol Set (PPS): Refers to the subgroup of treatment population who completes the trial and excluded the population that seriously violates the protocol (which means that study subjects violating the inclusion criteria or meeting exclusion criteria, loss to follow-up during the trial, cross enrollment, out-of-specification use of investigational products, out-of-window time, etc.).

Safety Set (SS): Set of all subjects who participate in the study and use the investigational products and undergo at least one safety evaluation after baseline. (The definitions of SS and FAS are the same. Therefore, SS is not defined separately).

Actual Treatment Set (ATS): All patients who participate in the randomized grouping, complete the trial, actually receive the scheduled treatment in the study (not necessarily consistent with the results of randomized grouping) and do not seriously violates the protocol. On the basis of PPS, only cross-enrolled patients are included, but they are then grouped and analyzed according to their actual treatment, i.e., the actual treatment set is formed.

The primary efficacy analysis will be based on FAS, PPS and ATS (if applicable). All baseline demographic data and secondary efficacy indicator analysis will be performed on the basis of FAS, and the safety evaluation will be performed on the basis of FAS.

# 6.4 Detailed rules for determination of analysis population set and flow chart

- (1) No investigational device is implanted: Subjects obtain random numbers but do not use any study-related treatment (implantation study group, control group or third party products);
- (2) Violation of inclusion and exclusion criteria: The subjects do not meet the inclusion criteria or meet the exclusion criteria set in the study protocol, and the violation of this protocol will seriously affect the results of primary efficacy endpoints; the sponsor, investigators and statisticians will jointly determine through a blind review meeting whether the protocol violation will seriously affect the results of primary efficacy endpoints;
- (3) Loss to follow-up during the trial: Subjects are unable to obtain the fracture union rate 24 weeks after the primary endpoint surgery;
- (4) Cross enrollment: Subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;
- (5) Out-of-window time: The difference between the follow-up date at 24 weeks after primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and the violation of this protocol may seriously affect the results of primary efficacy endpoints; the sponsor, investigators and statisticians will jointly determine through a blind review meeting whether the protocol violation will seriously affect the results of primary efficacy endpoints;
- (6) Out-of-specification use of investigational products: The specifications of the device implanted in the subject are not within the specification range specified in the study protocol;
- (7) Use of third party products: The subjects randomly assigned to the study group or the control group use third party products;

(8) FAS = Number of subjects enrolled in the trial - Number of subjects not implanted with any investigational device;

PPS = FAS - Number of subjects who seriously violate the study protocol;

ATS = PPS + Number of cross-enrolled subjects alone; ATS will be displayed if subjects are cross-enrolled in the trial, while ATS will not be displayed if no cross-enrollment occurs.

Number of subjects who seriously violate the study protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Out-of-window time + Out-of-specification use of investigational products + Use of third party products;

The priority of serious violations from study protocol: Loss to follow-up during the trial, cross enrollment, use of third party products, violation of inclusion and exclusion criteria, out-of-specification use of investigational products, out-of-window time; if the subjects meets the above two or more serious violations, the violations will be classified by priority;

Serious violations from study protocol in the statistical table can be listed according to the actual situation of the data. If the number of subjects who exceed the time window in both the study group and the control group is 0, then such information may not be shown in the table. Meanwhile, the list of subjects who are not implanted with any investigational device or have serious violations from study protocol will be provided, including site number, random number, gender, age, type, reason, FAS, PPS and ATS.



Figure 1 Flow chart for determination of analysis population data sets

## 6.5 Missing values, abnormal values and outlying values

For possible missing data in the study process, the missing of primary efficacy endpoints will be carried forward only in principle during the analysis. LOCF (Last Observation Carry Forward) was used as sensitivity analysis for the missing of primary efficacy endpoints. That is, the last observed value is used to replace the missing value. In the sensitivity analysis of the LOCF, the last observed value is "Nonunion of fracture" unless the fracture union is definitive. Other missing indicators will not be carried forward and will be directly analyzed based on the actually observed data.

Error and unreasonable data will be processed in the data cleaning process before statistical analysis. For withdrawal of subjects, this part of patient information will still be included in the final statistical analysis. Specific reasons for discontinuation or withdrawal of all patients will be explained in detail in the statistical report, and the missing primary endpoint due to early withdrawal will be analyzed according to the above strategy for processing missing values.

If the date (MMDDYYYY) of collection (non-CEC review data) during the trial is filled in with "UK" or "NA", no treatment will be done.

## 6.6 Significant level and statistical analysis software

For the primary endpoint, statistical analysis will be performed at the one-sided 0.025 significance level (corresponding to the one-sided confidence limit of the 95% confidence interval). For other endpoints, all statistical analysis will be performed at the two-sided 0.05 significance level (except for special instructions). SAS® 9.4 statistical software will be used for statistical analysis.

## 6.7 Site merging principle

This trial is to be conducted simultaneously in multiple clinical trial institutions, and the actual number of subjects successfully included in each site will vary. In order to avoid the influence of too few actual number of subjects successfully enrolled in the site on the stability and reliability of the primary endpoint analysis results, the sites with the actual number of subjects successfully enrolled less than 10 will be merged. According to previous experience and reference, site merging generally adopts the following two methods:

- (1) Sort the sites with the number of subjects actually enrolled less than 10 according to the site number, and merge the sites directly until the number of subjects in the sites is  $\geq 10$  after merging;
- (2) Merge the sites according to the principle of geographical proximity, and the number of subjects in the sites should be  $\geq 10$  after merging;

The site merging principle adopted in the statistical analysis will be further determined by the sponsor, the investigator and the statistician through a blind review meeting.

## 7. Statistical Analysis Indicators and Statistical Analysis Methods

# 7.1 Demographic indicators and other baseline indicators

Demographic data include gender, age, height, weight and BMI; other baseline indicators include the subject's medical history, SF-12v2 questionnaire, EQ-5D questionnaire and preoperative fracture status.

Version No.: V1.0

Where:

Age = (Date of informed consent - Date of birth)/ $\frac{365.25}{}$ ;

BMI = Body weight  $(kg)/(Height (m))^2$ .

The indicators in this part are mainly descriptive. Enumeration data are described by frequency and composition ratio, while measurement data are described by mean, standard deviation, median, quartile, maximum and minimum. The likelihood ratio Chi-square test will be used to compare the enumeration data between groups. Fisher's exact probability test will be used when the theoretical frequency in the fourfold table is less than 5.

## 7.2 Intraoperative information

The intraoperative information includes the subject's operation time, blood loss volume, blood transfusion volume, investigational device use, intraoperative fracture, etc.

The indicators in this part are mainly descriptive. Statistical analysis methods are the same as those in 7.1.

## 7.3 Primary endpoint

## The primary endpoint is the fracture union rate 24 weeks after surgery.

Fracture union success is a composite endpoint; in order for an individual subject's surgery implanted with TFNA or PFNA-II to be considered successful he/she must satisfy all of the following criteria:

- 1. No focal tenderness or lengthwise percussion pain, or abnormal movement
- 2. The frontal/lateral X-ray examination shows the vague or no fracture gap, or the continuous callus passing across the fracture line
- 3. No deformation or breakage is found in the investigational product

Calculation principle: Based on the postoperative 24-week follow-up of the fracture status and the X-ray examination results of the fracture site, the calculation principle is as follows:

- 1. It is determined as 'Yes' when the focal tenderness, lengthwise percussion pain and abnormal activity at the postoperative 24-week follow-up of the fracture are filled as 'NA', 'NA' and 'No', respectively;
- 2. It is determined as 'Yes' when the X-ray examination at the fracture site 24 weeks after surgery shows that the fracture line is 'vague' or 'disappeared'; or that the frontal/lateral X-ray examination shows the continuous callus passing across the fracture line is filled as 'Yes';
- ③. It is determined as 'Yes' when the X-ray examination at the fracture site 24 weeks after surgery shows that the implant is filled as 'good';

If ①, ② and ③ are determined as 'Yes', then the successful fracture union 24 weeks after surgery is determined as 'Yes'; if one of them is missing, it is determined as missing, that is, 'loss to follow-up during the trial'; others are determined as 'No';

For the primary endpoint, the analysis bases on the actual data (except missing data). LOCF (Last Observation Carry Forward) was used as sensitivity analysis for the missing of primary efficacy endpoints. The below 2 analysis tests will be used for the above analysis, and estimates of the differences in efficacy between the groups and bilateral two-sided 95% confidence interval will be given:

(1) CMH chi-square test with adjusted central effects;

Calculation method for non – inferiority P value:

Se=( Rate difference 95% upper limit of confidence interval - Rate difference 95% low limit of confidence interval)/2/ probit (1-0.05/2);

Z=( Investigational group-control group of difference in fracture union rates-non-inferiority margin)/Se;

P value=1-probnorm(Z);

Continuous correction Newcombe-Wilson for non-adjusted central; (2)

The result from test (1) will used for the primary analysis result, the result from test (2) will be used as sensitivity analysis result. If the lower limit of the bilateral two-sided 95% confidence interval on differences in efficacy between the study group and the control group (equal to the lower limit of unilateral 95% confidence interval) is greater than -10%, it can be considered that the investigational product is not inferior to the control product

If the actual study results show that other baseline variables (such as age and gender) are significantly different between the study group and the control group, it will be fully communicated to the investigator in the data analysis stage. Based on the results of univariate analysis for baseline variables and primary endpoint, previous literature references and the clinical expert experience, the indicators affecting the primary endpoint to cause imbalance between groups, i.e., confounding factors, will be further specified. These indicators will be considered into the generalized linear model for correction and included into the sensitivity analysis of the primary endpoint analysis.

## 7.4 Secondary endpoints

Secondary endpoints include the safety and effectiveness results, imaging outcomes and adverse events.

Adverse events (type and frequency) for all adverse events will be (1) compared for the study and control groups Version No.: V1.0

Calculation principle: Based on the collected adverse events in the CRF, if the subject has had at least one adverse event, it will be regarded as 'Yes'; otherwise, it will be 'No'.

The indicators in this part are mainly descriptive. Statistical analysis methods are the same as those in 7.1.

(2) 24-week revision rate, where revision is defined as any component removal for any reason.

Calculation principle: Based on the collected adverse events in the CRF, if the measure taken for the implant is filled as "Revision" and the difference between the date of occurrence of the event and the date of the operation is ≤196 days, the revision is determined as "Yes"; if postoperative 24-week follow-up is failed, it is determined as "Missing"; others are determined as 'No';

The indicators in this part are mainly descriptive. Statistical analysis methods are the same as those in 7.1.

(3) 24-week re-operation rate, where re-operation is defined as secondary operation of the fracture site for any reason.

Calculation principle: According to the AEs in CRF. If AE "re-operation" site collected in the CRF and occurrence of the event and the date of the operation is ≤196 days, it is determined as 'Yes'; if postoperative 24-week follow-up is failed, it is determined as 'Missing'; others are determined as 'No'.

The indicators in this part are mainly descriptive. Statistical analysis methods are the same as those in 7.1.

- (4) Clinical outcomes
- > SF-12
- > Harris Hip Score
- ➤ EQ-5D

# **Calculation principle for SF-12 Score:**

SF-12 v2 Questionnaire (each item consists of 8 parts: body functions, physical conditions, body pain, general health, mental health, emotional conditions, social functions and vitality) and general physical and mental health assessment.

Calculation principle: SF-12 scores will be calculated by special software, and statistical analysis will be performed using "NBS" variable.

The indicators in this part are mainly descriptive. The descriptive analysis results of the SF-12 score and the change from baseline at each follow-up will be given. The statistical analysis method is the same as 7.1. At the same time, the 95% confidence interval of the mean value of change value from each group, the

difference between groups and its 95% confidence interval are also provided.

## Calculation principle for Harris hip score:

Total Harris hip score: It can be calculated by adding the scores of each sub-item.

# (I) Regarding the complaint pain score (44 points in total), the specific points are as follows:

None, or ignores it (44 points)

Slight, occasional, no compromise in activities (40 points)

Mild pain, no effect on average activities (30 points)

Moderate pain, tolerable (20 points)

Marked pain, serious limitation of activities (10 points)

Totally disabled, crippled, pain in bed, bedridden (0 point)

# (II) Function score (47 points in total): Gait score (33 points) + daily life score (14 points), the specific points are as follows:

## Gait score (33):

- ① Support: None (11 points); Cane for long walks (7 points); Cane most of time (5 points); One crutch (3 points); Two canes (2 points); Two crutches or not able to walk (0 point)
- ② Distance Walked: Unlimited (11 points); Six blocks (30 minutes) (8 points); Two or three blocks (10 or 15 minutes) (5 points); Indoors only (2 points); Bed and chair only (0 point)
- ③ Limp: None (11 points); Slight (8 points); Moderate (5 points); Severe or unable to walk (0 point)

## Daily life score (14 points):

- ① Put on Shoes and Socks: With ease (4 points); With difficulty (2 points); Unable (0 point)
- ② Stairs: Normally without using a railing (4 points); Normally using a railing (2 points); In any manner (1 point); Unable to do stairs (0 point)
- ③ Enter public transportation: Yes (bus) (1 point); No (bus) (0 point)
- ④ Sitting: Comfortably in ordinary chair for one hour (5 points); On a high chair for 30 minutes (3 points); Unable to sit comfortably in any chair (0 point)

# (III) Physical sign score (4 points in total), the specific points are as follows:

Whether all of the following conditions exist: (Less than 30° fixed flexion contracture; Less than 10° fixed internal rotation in extension; Less than 10° fixed

abduction; Limb length discrepancy less than 3.2 cm (1.5 inches);)

Yes (4 points), No (0 point)

- (IV) Physical examination score: Score result = The sum of A, B, C and D divided by 20; the specific points are as follows (refer to computation rule for Harris Hip Score in <a href="http://www.orthopaedicscores.com">http://www.orthopaedicscores.com</a>, which was approved by the Journal of Bone & Joint Surgery):
- A. Total flexion: None (0 point), 0 >8 (0.4 points), 8 >16 (0.8 points), 16 >24 (1.2 points), 24 >32 (1.6 points), 32 >40 (2 points), 40 >45 (2.25 points), 45 >55 (2.55 points), 55 >65 (2.85 points), 65 >70 (3 points), 70 >75 (3.15 points), 75 >80 (3.3 points), 80 >90 (3.6 points), 90 >100 (3.75 points), 100 >110 (3.9 points);
- B. Total abduction: None (0 point), 0 > 5 (0.2 points), 5 > 10 (0.4 points), 10 > 15 (0.6 points), 15 > 20 (0.65 points);
- C. Total external rotation: None (0 point), 0 > 5 (0.1 point), 5 > 10 (0.2 points), 10 > 15 (0.3 points);

Total internal rotation: None (0 point), 0 > 5 (0.05 points), 5 > 10 (0.1 points), 10 > 15 (0.15 points);

Total Harris hip score: It can be calculated by adding the scores of the above four sub-items.

- If a sub-score is missing then the total score cannot be calculated
- If total score exceeds 100 then it should be forced to be 100

The indicators in this part are mainly descriptive. The descriptive analysis results of Harris hip score at each follow-up will be given. The statistical analysis method is the same as 7.1.

## **EQ-5D** questionnaire:

Based on the EQ-5D questionnaire collected in the CRF, the analysis results of subjects' health status and health index are given. The analysis results 12 and 24 weeks after surgery are given, respectively.

## **Calculation principle:**

Health status is measured in five dimensions (activity level, self-care, daily activities, pain/discomfort, anxiety/depression). Each dimension contains five levels: no difficulty, mild difficulty, moderate difficulty, severe difficulty, and extreme difficulty (marked 1-5). The health status of each subject is determined by arranging the five dimensions of each subject.

Health index is calculated by 《EQ-5D-5L Crosswalk Index Value Calculator.v2.xls》.

The indicators in this part are mainly descriptive. A descriptive analysis of each follow-up health index and changes relative to baseline will be presented. Statistical analysis methods are the same as those in 7.1.

(5) Radiographs: incidence of complications such as loosening or cut-out that require reoperation or revision.

Calculation principle: Based on the adverse events collected in the CRF. If the measure taken for the implant is filled as "Revision" or AE "re-operation" collected in the CRF, it is determined as 'Missing'; otherwise are determined as 'No'

The indicators in this part are mainly descriptive. Statistical analysis methods are the same as those in 7.1.

## 7.5 Follow-up data

The follow-up data include the frontal/lateral X-ray examination of fracture sites 1 week, 6 weeks, 12 weeks and 24 weeks after surgery, SF-12v2 health assessment scale, EQ5D and Harris hip score.

For indicators related to follow-up data, descriptive analysis is mainly performed. Statistical analysis methods are the same as those in 7.1.

## 7.6 Laboratory examinations

Laboratory test indicators include complete blood count and blood biochemical test. Blood test includes white blood cell (WBC), neutrophil percentage, red blood cell (RBC), hemoglobin, platelet, international normalized ratio (INR) and activated partial thromboplastin time (APTT); blood biochemical test includes alanine aminotransferase (ALT), aspartate aminotransferase (AST), albumin (ALB), cholesterol (CHOL), triglyceride (TRIG), creatinine (CREA), blood urea nitrogen (BUN), urea (UREA), uric acid (UA), low density lipoprotein (LDL-C), high-density lipoprotein (HDL-C), blood glucose (GLU), C-reactive protein (CRP) and hypersensitive CRP.

As for the laboratory examination indicators, the outcomes immediately after surgery relative to the preoperative conditions will be given. There are mainly five cases listed, including "Normal  $\rightarrow$  Abnormal (with clinical significance)", "Normal  $\rightarrow$  Abnormal (without clinical significance)", "Normal  $\rightarrow$  Normal", "Abnormal  $\rightarrow$  Abnormal"; the descriptive analysis method is mainly adopted. Statistical analysis methods are the same as those in 7.1. Meanwhile, the list of subjects presenting "Normal  $\rightarrow$  Abnormal (with clinical significance)" will be given, including laboratory examination indicators, site number, random number, group, age, gender, and laboratory indicator test values before surgery and immediately after surgery.

## 7.7 Concomitant medication, adverse events (AEs) or serious adverse events

## (SAEs)

For concomitant medication, the subject's concomitant medication is provided in the form of a list.

The AEs and investigational device-related AEs in subjects will be tabulated and summarized, respectively. The list of subjects reported with AEs/ investigational device-related AEs includes site number, random number, group, age, gender, name of AE (SOC code), name of AE (PT code), time of postoperative occurrence (day), remission time (day), severity, measures taken, outcome, correlation with surgery, correlation with investigational device, withdrawal from the trial due to AEs, whether it is unanticipated adverse device effect (UADE), device failure or SAE.

Investigational device-related AEs refer to those "definitely related", "probably related" and "possibly related" with the investigational device;

Time of postoperative occurrence (day) = Date of occurrence of AE - Date of surgery,

Remission time (day) = End date of AE - Date of occurrence of AE.

The summary form will list the total number of cases of AEs/investigational device-related AEs, the total number of subjects suffering from AEs/investigational device-related AEs.

Wherein, the total case of AEs refers to the number of subjects suffering from AEs, and the AEs occur in the subject at least one time, which is considered as "Yes";

Statistical analysis of the severity of adverse events, the relationship with the study device and the relationship with the surgery was performed. If multiple adverse events occurred in a patient, the analysis was performed with the most severe or highest correlation.

The SAEs and investigational device-related SAEs in subjects will be tabulated and summarized, respectively; such data will be presented in the same form as AEs. The list of subjects reported with SAEs/investigational device-related SAEs includes site number, random number, group, age, gender, name of SAE (SOC code), name of SAE (PT code), time of postoperative occurrence (day), remission time (day), severity, outcome, correlation with surgery, correlation with investigational device and SAE.

The list and summary of UADEs in subjects will be presented respectively in the same form as AEs.

The calculation method of the time of postoperative occurrence (day) and remission time (day), the presentation of the summary form and the statistical principle are the same as those for AEs.

## 8. Generation of Statistical Graphs, Tables and Lists



Figure 1 Flow chart for determination of analysis population data sets

 Table 1
 Determination of analysis population

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2. Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 2 List of subjects who withdrawal the informed consent or seriously violate the protocol

| Site<br>No. | Random<br>No. | Group | Gender | Age | Type | Reason | FAS | PPS | ATS |
|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | | | | | |
| XXX | XXX | XXX | XXX | XXX | | | | | |

Note: If the subject is included in FAS, PPS and ATS, mark with " $\sqrt{}$ "; if the subject is not included in FAS, PPS and ATS, mark with " $\times$ ".

# Table 3 List of subjects who violate the protocol (CRF collection)

| Site No. | Random<br>No. | Group | Gender | Age | Туре | AE/SAE<br>related or<br>not | Withdrawal of subjects from the trial or not |
|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | | | ••••• |
| XXX | XXX | XXX | XXX | XXX | | | |

Table 4 Determination of analysis population in Beijing Jishuitan Hospital

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2. Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 5 Determination of analysis population in Peking University Third Hospital

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 6 Determination of analysis population in Chinese PLA General Hospital

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 7 Determination of analysis population in the Second Affiliated Hospital of Zhejiang University School of Medicine

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 8 Determination of analysis population in Shanghai General Hospital

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 9 Determination of analysis population in Nanfang Hospital Of Southern Medical University

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 10 Determination of analysis population in Affiliated Hospital of Nantong University

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);
Table 11 Determination of analysis population in West China Hospital, Sichuan University

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 12 Determination of analysis population in the First Affiliated Hospital of Guangzhou University of Chinese Medicine

| Indicator | Study group | Control group |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 13 Determination of analysis population in the University of Hong Kong - Shenzhen Hospital

| Indicator Study group | Control group | |
|---|---|---|
| Randomization | XXX (XX.X%) | XXX (XX.X%) |
| No investigational device is implanted | XXX (XX.X%) | XXX (XX.X%) |
| Serious protocol violation | | |
| Violation of inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Loss to follow-up during the trial | XXX (XX.X%) | XXX (XX.X%) |
| Cross enrollment | XXX (XX.X%) | XXX (XX.X%) |
| Use of third party products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-specification use of investigational products | XXX (XX.X%) | XXX (XX.X%) |
| Out-of-window time | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |
| ATS | XXX (XX.X%) | XXX (XX.X%) |

- 1. FAS = Number of subjects enrolled randomly Number of subjects not implanted with any investigational device;
- 2: Number of subjects who seriously violate the protocol = Violation of inclusion and exclusion criteria + Loss to follow-up during the trial + Cross enrollment + Use of third party products + Out-of-specification use of investigational products + Out-of-window time;
- 3. PPS = FAS Number of subjects who seriously violate the protocol; ATS = PPS + Number of cross-enrolled subjects alone;
- 4. No investigational device is implanted means that the subject has been given a random number but has not received any study-related treatment;

Loss to follow-up during the trial refers to the situation in which the fracture union rate 24 weeks after the primary endpoint surgery is not available;

Cross enrollment refers to the situation in which subjects randomly assigned to the study group receive the control products, while subjects randomly assigned to the control group receive the investigational products;

Out-of-specification use of investigational products refers to the situation in which the specification of the device implanted in the subject is not within the specification range specified in the study protocol;

Use of third party products refers to the situation in which the subjects randomly assigned to the study group or the control group use third party products;

Out-of-window time refers to the situation in which the difference between the follow-up date at 24 weeks after subjects have received the primary endpoint surgery and the surgery date do not fall within the range of [140, 196], and this protocol violation may seriously affect the results of primary efficacy endpoints;

5: Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 14 Statistical analysis results of subjects' demographic data

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Age (years) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Gender | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Male | XXX (XX.X%) | XXX (XX.X%) | | |
| Female | XXX (XX.X%) | XXX (XX.X%) | | |
| Marital status | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Married | XXX (XX.X%) | XXX (XX.X%) | | |
| Unmarried | XXX (XX.X%) | XXX (XX.X%) | | |
| Nationality | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Han nationality | XXX (XX.X%) | XXX (XX.X%) | | |
| Others | XXX (XX.X%) | XXX (XX.X%) | | |
| Job nature | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Manual worker | XXX (XX.X%) | XXX (XX.X%) | | |
| Non-manual worker | XXX (XX.X%) | XXX (XX.X%) | | |
| Retired | XXX (XX.X%) | XXX (XX.X%) | | |
| Unemployed | XXX (XX.X%) | XXX (XX.X%) | | |
| Incompetent | XXX (XX.X%) | XXX (XX.X%) | | |
| Others | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Age = (Date of informed consent Date of birth)/365.25;
- 5. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 15 Statistical analysis results of subjects' height and body weight

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Body weight (kg) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX<br>( XXX)X.XXXX | X.XXXX | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Height (cm) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| BMI(kg/m^2) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. BMI= Body weight (kg)/Height (m)2;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 16 Statistical analysis results of subjects' previous and current medical history

| Indicator | Indicaton | C4., J | Cont1 - | C+-+: | D 1 |
|---|---|---|---|---|---|
| Number of subjects (N miss) | Indicator | Study group | Control group | Statistics | P value |
| Yes XXX<br>(XXX%)<br>(XXX%) XXX<br>(XXXX%) XXX<br>(XXXXX) Still persist Number of subjects (N miss) XXX (XXXX)<br>(XXXX%) XXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | - | VVV ( VVV) | VVV ( VVV) | vvvvv | vvvv |
| No | 2 , | | , , | Α.ΧΧΧΧ | Α.ΑΑΑΑ |
| No | Yes | | $\lambda\lambda\lambda\lambda$ ( $\lambda\lambda.\lambda\%$ ) | | |
| Still persist | No | | XXX (XX X%) | | |
| Number of subjects (N miss) | NO | | AAA(AA.A/0) | | |
| Number of subjects (N miss) | Still persist | (111.2170) | | | |
| Yes XXX<br>(XX,X%)<br>(XX,X%) XXX (XX,X%)<br>(XX,X%) XXX (XX,X%) XXX (XX,X%) Malnutrition Number of subjects (N miss) XXX (XXX) XXX (XX,X%) XXXX (XX,X%) None XXX (XX,X%) XXX (XX,X%) XXXX (XX,X%) Ca XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) P XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Protein XXX (XX,X%) XXX (XX,X%) XXX (XX,X%) Others XXX (XX,X%) XXX (XX,X%) XXXX (XX,X%) Others XXX (XX,X%) XXXX (XX,X%) XXXX (XX,X%) Yes XXX (XX,X%) XXXX (XX,X%) XXXXX (XX,X%) No XXX (XX,X%) XXXX (XX,X%) XXXXX (XX,XX) Yes XXX (XX,X%) XXXX (XX,XX) XXXXX (XX,XX) Yes XXX (XX,X%) XXXX (XX,XX,X%) XXXXX (XX,XX) No XXX (XX,X%) XXXX (XX,XX,X%) XXXXX (XX,XX,XX) No XXX (XX,X%) XXXX (XX,XX,XX,XX) XXXXX (XX,XX,XX,XX,XX,XX,XXXX Yes XXX (XX,XX,XX,XX,XX,XX,XX,XX,XX,XX,XX,XX,XX, | _ | XXX (XXX) | XXX (XXX) | x xxxx | X XXXX |
| No | 2 , | ` ' | ` ' | 71.71717171 | 71.71717171 |
| No XXX<br>(XX.X%) XXX (XX.X%) Malnutrition Number of subjects (N miss) XXX (XXX) XXX (XXXX) XXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | 105 | | 71711 (7171.7170) | | |
| Malnutrition | No | , , | XXX (XX.X%) | | |
| Malnutrition Number of subjects (N miss) XXX (XXX) XXXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | () | | |
| Number of subjects (N miss) | Malnutrition | , | | | |
| None | | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Ca | 2 , | • • • | , , | | |
| P | | | , | | |
| Protein | Ca | XXX | XXX (XX.X%) | | |
| Protein | | (XX.X%) | , , | | |
| Protein XXX<br>(XX.X%)<br>(XX.X%) XXX<br>XXX (XX.X%) Others XXX<br>XXX<br>(XX.X%) XXX (XX.X%) Still persist XXX<br>(XX.X%) XXX (XXX)<br>XXX (XXXX) XXXX (XXXX)<br>XXX (XXXX%) No XXX<br>(XX.X%) XXX (XXXX%) Anemia XXX (XXXX)<br>XXX (XXXXX) XXXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | P | XXX | XXX (XX.X%) | | |
| Comparison of Subjects (N miss) XXX (XXX) XXX (XXXX) XXXX (XXXX XXXX | | (XX.X%) | | | |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Protein | | XXX (XX.X%) | | |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | | (XX.X%) | | | |
| Others XXX<br>(XX.X%) XXX (XX.X%) Still persist XXX (XXX) XXX (XXX) XXXX (XXXX) XXXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Fe | | XXX (XX.X%) | | |
| (XX.X%) Still persist Number of subjects (N miss) XXX (XXX) XXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | |
| Still persist | Others | | XXX (XX.X%) | | |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | ~ *** | (XX.X%) | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | - | | | | |
| No | 2 , | • • • | , , | X.XXXX | X.XXXX |
| No XXX<br>(XX.X%) XXX (XX.X%) Anemia Number of subjects (N miss) XXX (XXX) XXX (XXX) X.XXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes | | XXX (XX.X%) | | |
| Anemia | N | | 3/3/3/ (3/3/ 3/0/) | | |
| Anemia $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | No | | XXX (XX.X%) | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | A | $(\Lambda\Lambda.\Lambda\%0)$ | | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | | VVV ( VVV) | VVV ( VVV) | VVVVV | VVVVV |
| No $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | - · | | , , | Α.ΧΧΧΧ | Α.ΧΧΧΧ |
| No $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Yes | | XXX(XX.X%) | | |
| $(XX.X\%) \\ Still persist \\ Number of subjects (N miss) & XXX (XXX) & XXX (XXX) & X.XXXX & X.XXXX \\ Yes & XXX & XXX (XX.X\%) & XXX (XX.X\%) \\ No & XXX & XXX (XX.X\%) & XXX (XX.X\%) \\ Hormone deficiency & XXX (XXX) & XXX (XXX) & X.XXXX & X.XXXX \\ Number of subjects (N miss) & XXX (XXX) & XXX (XXX) & X.XXXX & X.XXXX \\ None & XXX & XXX (XXX.X\%) & X.XXXX & X.XXXXX \\ Medical Research & Biometrics Center, National & Version No.: V1.0 & 41/129 \\ \end{bmatrix}$ | No | | VVV (VV V0/) | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | INO | | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda\%)$ | | |
| Number of subjects (N miss) XXX ( XXX ) XXX ( XXX ) X.XXXX XXXXXX Yes XXX XXX ( XXX ) XXX ( XXXX ) XXXXXX XXXXXX XXX ( XXX ) XXX ( XXX ) XXX ( XXX ) XXX ( XXX ) XXX ( XXX ) XXX ( XXX ) XXXX XXXXX XXXXX XXXXX XXXXX XXXXX | Still persist | $(\Lambda\Lambda.\Lambda/0)$ | | | |
| $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | _ | VVV ( VVV) | VVV ( VVV) | v vvvv | v vvvv |
| $(XX.X\%) \\ No \\ XXX \\ (XX.X\%) \\ Hormone deficiency \\ Number of subjects (N miss) \\ XXX (XXX) \\ XXX (XXX) \\ XXX (XXX) \\ XXX (XXX) \\ XXX (XXXX) \\ XXX (XXXX) \\ XXX (XXXXX) \\ XXX (XXXXXXXXXX$ | - · | * * | ` ' | Α.ΑΑΑΑ | Α.ΑΑΑΑ |
| No $ \begin{array}{ccccccccccccccccccccccccccccccccccc$ | 1 CS | | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| Hormone deficiency $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | No | | XXX (XX X%) | | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | 140 | | AAA(AA.A/0) | | |
| Number of subjects (N miss) XXX ( XXX) XXX ( XXX) XXXXXX XXXXX XXXXX XXXXX XXXXX XXXXX XXXX | Hormone deficiency | (12121170) | | | |
| None $ \begin{array}{ccc} XXX & XXX (XX.X\%) \\ (XX.X\%) & & & & & & & \\ & & & & & & \\ & & & & & \\ & & & & & & \\ & & & & & & \\ & & & & & & \\ & & & & & \\ & & & & & \\ & & & & \\ & & & \\ & & & & \\ & & & & \\ & & & \\ & & & & \\ & & & \\ & & & & \\ & & & \\ & & & \\ & & & & \\ & & \\ & & & \\ &$ | | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $(XX.X\%) \label{eq:continuous} $ Medical Research & Biometrics Center, National | 2 , | | , , | | |
| Medical Research & Biometrics Center, National Version No.: V1.0 41/129 | 1,0110 | | 2222 (222271/0) | | |
| | Medical Research & Biometrics Center. Nati | ` , | Version No.: V1.0 | l | 41/129 |
| | | | | | · <b></b> |

| Growth hormone | XXX<br>(XX.X%) | XXX (XX.X%) | | |
|-----------------------------|----------------|-------------|--------|--------|
| Parathyroid hormone | XXX<br>(XX.X%) | XXX (XX.X%) | | |
| Others | XXX<br>(XX.X%) | XXX (XX.X%) | | |
| Still persist | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX<br>(XX.X%) | XXX (XX.X%) | | |
| No | XXX<br>(XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 16 Statistical analysis results of subjects' previous and current medical history (continued 1)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Diabetes mellitus | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes (satisfactory control) | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes (unsatisfactory control) | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Allergic history | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Other complications | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Still persist | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Smoke within one year or not | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Number of cigarettes/day | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Still persist | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Drink within one year or not | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 16 Statistical analysis results of subjects' previous and current medical history (continued 2)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| ml/day | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Still persist | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Surgical history | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 17 Statistical analysis results of subjects' preoperative SF-12v2 questionnaire

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (body functions) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| SF-12 score (physical conditions) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm\! XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| SF-12 score (body pain) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm\! XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| SF-12 score (general health) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| SF-12 score (vitality) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm\! XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| SF-12 score (social functions) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 17 Statistical analysis results of subjects' preoperative SF-12v2 questionnaire (continued)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (emotional conditions) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| SF-12 score (mental health) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| SF-12 score (total physical health sco | ore) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| SF-12 score (total mental health score | e) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 18 Statistical analysis results of subjects' preoperative EQ-5D questionnaire

| | <u>luestionnaire</u> | | | |
|---|---|---|---|---|
| Indicator | Study group | Control group | Statistics | P value |
| Activity level | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Walk easily | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to walk | XXX (XX.X%) | XXX (XX.X%) | | |
| Self-care | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Daily activities (such as work, study, house | work, family or ent | ertainment) | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Pain/discomfort | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Anxiety/depression | , | , , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |

Notes:

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.

- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 18 Statistical analysis results of subjects' preoperative EQ-5D questionnaire (continued)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Health index | | | | |
| Number of subjects (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 19 Statistical analysis results of subjects' preoperative fractures

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Limb malformation | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Flexion | XXX (XX.X%) | XXX (XX.X%) | | |
| Shortening | XXX (XX.X%) | XXX (XX.X%) | | |
| Limb malformation and external rotat | ion | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| External rotation < 30° | XXX (XX.X%) | XXX (XX.X%) | | |
| 30° < External rotation < 60° | XXX (XX.X%) | XXX (XX.X%) | | |
| External rotation≥60° | XXX (XX.X%) | XXX (XX.X%) | | |
| Closed fracture | , | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| C 0 | XXX (XX.X%) | XXX (XX.X%) | | |
| CI | XXX (XX.X%) | XXX (XX.X%) | | |
| CII | XXX (XX.X%) | XXX (XX.X%) | | |
| C III | XXX (XX.X%) | XXX (XX.X%) | | |
| Open fracture | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| O | I | XXX (XX.X%) | XXX<br>(XX.X%) | |
| O II | XXX (XX.X%) | XXX (XX.X%) | , | |
| O III | XXX (XX.X%) | XXX (XX.X%) | | |
| O IV | XXX (XX.X%) | XXX (XX.X%) | | |
| Degree of limb swelling | , | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mild | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 20 Statistical analysis results of subjects' x-ray examination before surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Fracture site - Lower limbs | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Left | XXX (XX.X%) | XXX (XX.X%) | | |
| Right | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of trochanteric fracture | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Simple pertrochanteric fracture (31-A1) | XXX (XX.X%) | XXX (XX.X%) | | |
| Comminuted pertrochanteric fracture (31-A2) | XXX (XX.X%) | XXX (XX.X%) | | |
| Intertrochanteric fracture (31-A3) | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of fracture | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Open | XXX (XX.X%) | XXX (XX.X%) | | |
| Closed | XXX (XX.X%) | XXX (XX.X%) | | |
| Reason for fracture | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| High energy damage (such as, MVA) | XXX (XX.X%) | XXX (XX.X%) | | |
| Low energy damage (such as, a fall in a standing position) | XXX (XX.X%) | XXX (XX.X%) | | |
| Others | XXX (XX.X%) | XXX (XX.X%) | | |
| Whether there are other fractures or no | ot | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 21 Statistical analysis results of subjects' use of investigational devices

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Intramedullary nails - Product No. | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| Head elements - Product No. | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| Whether to implant distal locking screen | ews | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Distal locking screws - Product No. | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| ļ | | | | |
| Whether to implant proximal locking | screws | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Proximal locking screws - Product No | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| l | | | | |
| Whether to implant intermediate lock | • | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 21 Statistical analysis results of subjects' use of investigational devices (continued)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Intermediate locking screws - Produc | t No. | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| End caps - Product No. | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |
| XXXXX | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 22 Statistical analysis results of subjects' use of other devices

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Any other internal or external fixatio | n is used at the same t | ime | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site of application | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Femur | XXX (XX.X%) | XXX (XX.X%) | | |
| Tibia and fibula | XXX (XX.X%) | XXX (XX.X%) | | |
| Ulna and radius | XXX (XX.X%) | XXX (XX.X%) | | |
| Humerus | XXX (XX.X%) | XXX (XX.X%) | | |
| Others | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 23 Statistical analysis results of subjects' surgical details

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Surgery time (hour) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Intraoperative blood loss volume (ml | L) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Intraoperative blood transfusion volu | ime (mL) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Specific components of intraoperative | e blood transfusion | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Concentrated red blood cell | XXX (XX.X%) | XXX (XX.X%) | | |
| Whole blood | XXX (XX.X%) | XXX (XX.X%) | | |
| Platelet | XXX (XX.X%) | XXX (XX.X%) | | |
| Fresh frozen plasma (FFR) | XXX (XX.X%) | XXX (XX.X%) | | |
| Others | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 24 Statistical analysis results of subjects' intraoperative fractures

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Closed fracture | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| C 0 | XXX (XX.X%) | XXX (XX.X%) | | |
| CI | XXX (XX.X%) | XXX (XX.X%) | | |
| CII | XXX (XX.X%) | XXX (XX.X%) | | |
| CIII | XXX (XX.X%) | XXX (XX.X%) | | |
| Open fracture | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 0 | I | XXX (XX.X%) | XXX<br>(XX.X%) | |
| O II | XXX (XX.X%) | XXX (XX.X%) | | |
| O III | XXX (XX.X%) | XXX (XX.X%) | | |
| O IV | XXX (XX.X%) | XXX (XX.X%) | | |
| Degree of limb swelling | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mild | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe | XXX (XX.X%) | XXX (XX.X%) | | |
| Whether there is vascular injury? | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Whether there is nerve injury? | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Volume of drainage 24 hours after s | urgery (mL) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Method for reduction of fracture | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Closed reduction | XXX (XX.X%) | XXX (XX.X%) | | |
| Open reduction | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 24 Statistical analysis results of subjects' intraoperative fractures (continued)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Reaming | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Not reamed | XXX (XX.X%) | XXX (XX.X%) | | |
| Reamed | XXX (XX.X%) | XXX (XX.X%) | | |
| Diameter after reaming (mm) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Incision closure | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Tension-free suture | XXX (XX.X%) | XXX (XX.X%) | | |
| Tension suture | XXX (XX.X%) | XXX (XX.X%) | | |
| Non-direct closure | XXX (XX.X%) | XXX (XX.X%) | | |
| Whether there is device-related even | t | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 3. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 25 Statistical analysis results of subjects' evaluation on product operability and tools during the surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Difficulty level of determining the na | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Average | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficulty level of inserting an intram | , | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Average | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficulty level of proximal locking | · · · · · · | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Average | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficulty level of distal locking | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Average | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficulty level of placing end caps | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Average | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Whether the placement of intramedul | lary nails has an impa | act on restoration | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No impact | XXX (XX.X%) | XXX (XX.X%) | | |
| Better than before | XXX (XX.X%) | XXX (XX.X%) | | |
| Worse than before | XXX (XX.X%) | XXX (XX.X%) | | |
| Instrument and its quantity | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Average | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Tools in the toolbox | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Average | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |

Notes:

<sup>1.</sup> The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;

<sup>2.</sup> Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 26 Statistical analysis results of subjects' intraoperative AEs

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether there are adverse events or c | complications in the s | subjects during the su | rgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 27 Statistical analysis results of subjects' intraoperative medication records

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new drugs are added to the medication is changed | concomitant medicat | ion or whether the or | iginal concom | itant |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 28 Statistical analysis results of subjects' intraoperative combination therapy

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new types of combination the | herapy are added | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 29 (FAS) Primary endpoint - statistical analysis results of fracture union rate of subjects at each site 24 weeks after surgery

| Indicator | Study group | Control group | | P value |
|---|---|---|---|---|
| Site 01 Beijing Jishuitan Hospital - S | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 02 Peking University Third Hos | | ture union 24 weeks | after surgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 03 Chinese PLA General Hospit | * * | • | er surgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | · | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 04 The Second Affiliated Hospit | | • | ine - Successi | ful fracture |
| union 24 weeks after surgery | <u>-</u> J <i>g</i> | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 05 Shanghai General Hospital - | | • | urgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | , , | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 05 Nanfang Hospital of Southern | | • | union 24 wee | ks after |
| surgery | J | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 07 The First Affiliated Hospital | of Nantong University | • | e union 24 we | eks after |
| surgery | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 08 West China Hospital, Sichuai | * * | sful fracture union 24 | weeks after s | urgery |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 09 The First Affiliated Hospital union 24 weeks after surgery | | ` / | cine - Success | sful fracture |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | | 1 111 11 11 11 1 | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 10 University of Hong Kong - S | ` / | • | on 24 weeks a | fter |
| surgery | nonzhon 1105piun - 5u | | on 2 i woons a | .1.01 |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | 21.21/1/1/1 | 21.21/1/1/1 |
| 100 | ZXXXX (ZXZX.ZX/U) | 232323 (2323.23/U) | | |

Table 29 (FAS) Primary endpoint - statistical analysis results of fracture union rate of subjects at each site 24 weeks after surgery (continued)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| #1 merged site- Successful fracture u | nion 24 weeks after s | urgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. #1: hospital XXX, hospital XXX and hospital XXX merged;
- 2. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 30 (FAS) Primary endpoint - Statistical analysis results of subjects' fracture union rate 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Successful fracture union 24 weeks af | ter surgery <sup>#1</sup> | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| No | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Difference in success rate (study group - co | ontrol group) and 95% CI | XX.X% [ XX.X | %; XX.X%] | |
| P value in non-inferiori | ty test #3 | X.XXXX | | |
| Difference in success rate (study group - co | ontrol group) and 95% CI | XX.X% [ XX.X | %; XX.X%] | |
| P value in non-inferiori | ty test #4 | X.XXXX | | |
| Successful fracture union 24 weeks at | eter surgery <sup>#2</sup> | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | | |
| Yes | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| No | XXX (XX.X%) X | | | |
| Difference in success rate (study group - control group) and 95% CI | | XX.X% [ XX.X | %; XX.X%] | |
| P value in non-inferiority test #3 | | X.XXXX | - | |
| Difference in success rate (study group - control group) and 95% CI | | XX.X% [ XX.X | %; XX.X%] | |
| P value in non-inferiori | ty test #4 | X.XXXX | | |

1. #3 is analyzed by CMH chi-square test with adjusted sites, estimate the difference in success rate and non-inferiority test the P value;

#4 is analyzed by Continuous correction Newcombe-Wilson for non-adjusted central, estimate the difference in success rate and non-inferiority test the P value;

- 2. #1: The primary efficacy indicators of the subjects lost to follow-up during the trial were not processed;
- #2: The primary efficacy indicators of the subjects lost to follow-up during the trial were carried forward by LOCF;
- 3. If the lower limit of 95% CI of the difference in the rates of the study group and the control group is greater than the non-inferiority margin of -10%, then the investigational product is considered non-inferior to the control product, i.e., the non-inferiority conclusion is established in this trial.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 31 (PPS) Primary endpoint - statistical analysis results of fracture union rate of subjects at each site 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Site 01 Beijing Jishuitan Hospital - Su | accessful fracture unio | on 24 weeks after su | rgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 02 Peking University Third Hosp | ital - Successful fract | ure union 24 weeks | after surgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 03 Chinese PLA General Hospita | l - Successful fractur | e union 24 weeks aft | er surgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 04 The Second Affiliated Hospita union 24 weeks after surgery | al of Zhejiang Univer | sity School of Medic | ine - Success | ful fracture |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 05 Shanghai General Hospital - S | Successful fracture un | ion 24 weeks after si | urgery | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 05 Nanfang Hospital of Southern | ` ' | | union 24 wee | ks after |
| Surgery | VVV ( VVV) | VVV ( VVV) | VVVVV | VVVVV |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | 24 | alra aftan |
| Site 07 The First Affiliated Hospital osurgery | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX(XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 08 West China Hospital, Sichuan | University - Success | ful fracture union 24 | weeks after s | ~ , |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX(XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 09 The First Affiliated Hospital ounion 24 weeks after surgery | of Guangzhou Univers | sity of Chinese Medi | cine - Succes | sful fracture |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Site 10 University of Hong Kong - Sh | * * | | on 24 weeks a | fter |
| Surgery | VVV ( VVV) | VVV (VVV) | v vvvv | v vvvv |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

Table 31 (PPS) Primary endpoint - statistical analysis results of fracture union rate of subjects at each site 24 weeks after surgery (continued)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| #1 merged site- Successful fracture u | nion 24 weeks after s | urgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. #1: hospital XXX, hospital XXX and hospital XXX merged;
- 2. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 32 (PPS) Primary endpoint - Statistical analysis results of subjects' fracture union rate 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Successful fracture union 24 weeks a | after surgery | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Difference in success rate (study group - control group) and 95% CI XX.X% [XX.X%; XX.X%] P value in non-inferiority test #1 X.XXXX | | | | |
| Difference in success rate (study group - or P value in non-inferior | <b>U</b> 17 | CI XX.X% [ XX.X<br>X.XXXX | [%; XX.X%] | |

- 1. #1 is analyzed by CMH chi-square test with adjusted sites, estimate the difference in success rate and non-inferiority test the P value;
- #2 is analyzed by Continuous correction Newcombe-Wilson for non-adjusted central, estimate the difference in success rate and non-inferiority test the P value;
- 2. If the lower limit of 95% CI of the difference in the rates of the study group and the control group is greater than the non-inferiority margin of -10%, then the investigational product is considered non-inferior to the control product, i.e., the non-inferiority conclusion is established in this trial.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 33 (ATS) Primary endpoint - Statistical analysis results of subjects' fracture union rate 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Successful fracture union 24 weeks at | fter surgery | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Difference in success rate (study group - c | ontrol group) and 95% ( | <br>ΣΙ ΧΧ.Χ% [ ΧΧ.Σ | <br>ζ%; XX.Χ%] | |
| P value in non-inferiority test #1 | | X.XXXX | , | |
| Difference in success rate (study group - c | ontrol group) and 95% ( | CI XX.X% [ XX.X | X%; XX.X%] | |
| P value in non-inferiori | ty test #2 | X.XXXX | | |

- 1. #1 is analyzed by CMH chi-square test with adjusted sites, estimate the difference in success rate and non-inferiority test the P value;
- #2 is analyzed by Continuous correction Newcombe-Wilson for non-adjusted central, estimate the difference in success rate and non-inferiority test the P value;
- 2. ATS = PPS + The number of subjects with cross enrollment but without other serious violations of the study protocol.
- 3. If the lower limit of 95% CI of the difference in the rates of the study group and the control group is greater than the non-inferiority margin of -10%, then the investigational product is considered non-inferior to the control product, i.e., the non-inferiority conclusion is established in this trial.
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 34 (FAS) Secondary endpoint - Statistical analysis results of adverse events of subjects

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total number of AEs | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The total number of AEs refers to the number of subjects suffering from AEs, and the AEs occur in the subject at least one time, which is considered as "Yes".
- 2. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 35 (FAS) Secondary endpoint - Statistical analysis results of subjects' revision rate 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether revision is required 24 week | s after surgery | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 36 (FAS) Secondary endpoint - Statistical analysis results of subjects' re-operation rate 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether re-operation is required 24 w | eeks after surgery | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 37 (FAS) Secondary endpoint - Statistical analysis results of subjects' Harris hip score 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total Harris hip score | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);
Table 38 (FAS) Secondary endpoint - Statistical analysis results of subjects' Harris hip score 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total Harris hip score | | | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 39 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery

| · | | | | |
|---|---|---|---|---|
| Indicator | Study group | Control group | Statistics | P value |
| SF-12 score (body function | ns) | | | |
| Number of subjects | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| (N miss) | | | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (bo | dy functions) relative to b | efore surgery | | |
| Number of subjects | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| (N miss) | | | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| 95% confidence | (XX.XX, XX.XX) | (XX.XX,XXXXXX) | | |
| interval | | | | |
| The difference and | XX.XX(XX.XX,XX.X | X) | | |
| 95% confidence | | | | |
| interval | | | | |
| SF-12 score (physical cond | | | | |
| Number of subjects | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| (N miss) | | | | |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | XX.XX ±XX.XX | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (ph | • | | | |
| Number of subjects | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| (N miss) | 3/3/ 3/3/ +3/3/ 3/3/ | 3/3/ 3/3/ +3/3/ 3/3/ | | |
| Mean $\pm$ SD | XX.XX ±XX.XX | XX.XX ±XX.XX | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| 95% confidence | (XX.XX, XX.XX) | (XX.XX, XX.XX) | | |
| interval | | | | |
| | X.XX(XX.XX,XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |
| SF-12 score (body pain) | 3/3/3/ ( 3/3/3/) | 3/3/3/ ( 3/3/3/) | 37. 37373737 | 37 37373737 |
| Number of subjects | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| (N miss) | VV VV +VV VV | VV VV +VV VV | | |
| Mean ± SD | XX.XX ±XX.XX | XX.XX ±XX.XX | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| | | | , | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 39 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery (continued 1)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (general health) | | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (gene | eral health) relative to be | fore surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| 95% confidence interval | .XX(XX.XX, XX.XX) | | | |
| SF-12 score (vitality) | VVV ( VVV) | VVV ( VVV) | vvvvv | vvvvv |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (vital | ity) relative to before su | rgery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and XX 95% confidence interval | .XX(XX.XX, XX.XX) | | | |

Version No.: V1.0

74/129

Medical Research & Biometrics Center, National

Center for Cardiovascular Diseases

| SF-12 score (social functions) | | | | |
|---|---|---|---|---|
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm \! XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (social to | functions) relative to b | efore surgery | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence (X | X.XX,XX.XX) | (XX.XX,XX.XX) | | |
| interval | | | | |
| The difference and XX.X | X(XX.XX,XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 39 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery (continued 2)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (emotional con | | Condoi group | Statistics | 1 (4140 |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | | | |
| Minimum; maximum | XX.XX ;XX.XX | | | |
| Change in SF-12 score (emo | · · | ŕ | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and 95% confidence interval | X.XX(XX.XX,XX.XX) | | | |
| SF-12 score (mental health) | | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (men | · · | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| 95% confidence interval | X.XX(XX.XX,XX.XX) | | | |
| SF-12 score (total physical ) | · · | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Medical Research & Biometrics | Center, National | Version No.: | V1.0 | 76/129 |

Center for Cardiovascular Diseases

| Change in SF-12 score | total pl | hysical health s | score) relative to | before surgery |
|---|---|---|---|---|

| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
|---|---|---|---|---|
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence | (XX.XX, XX.XX) | (XX.XX,XX.XX) | | |

interval

The difference and XX.XX(XX.XX,XX.XX)

95% confidence

interval

Notes:

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 39 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery (continued 3)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (total mental health | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm \! XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (total me | ental health score) relat | tive to before surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| 95% confidence (2 interval | XX.XX ,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and 95% confidence interval XX.X | XX(XX.XX ,XX.XX) | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 40 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (body functions) | ) | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (body | | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Tylininani, maximani | 7171.7171 ,7171.7171 | 7171.7711 ,7171.7711 | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and 95% confidence interval | X.XX(XX.XX ,XX.XX) | | | |
| SF-12 score (physical condit | ions) | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (phys | | · · | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| | X.XX(XX.XX ,XX.XX) | | | |
| 95% confidence interval | A.AA(AA.AA ,AA.AA) | | | |
| SF-12 score (body pain) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Medical Research & Biometrics ( | | Version No.: V1 | 1.0 | 79/129 |
| interior resourch & Diometros | | , 5151011 1 to V 1 | | 171127 |

Center for Cardiovascular Diseases

| Change in SF-12 score (body pain) relative to before surgery | | | | |
|---|---|---|---|---|
| Number of subjects (miss) | N XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | n XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and 95% confidence interval | XX.XX(XX.XX,XX.XX) | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 40 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery (continued 1)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (general health) | | | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (general hea | alth) relative to befo | re surgery | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| 0.50/ 6.1 (3/3/ | 3/3/ 3/3/ 3/3/ | (3/3/ 3/3/ 3/3/ 3/3/ | | |
| 95% confidence (XX interval | .XX, XX.XX) | (XX.XX,XX.XX) | | |
| | vv vv vv vv | | | |
| 95% confidence | XX.XX ,XX.XX) | | | |
| interval | | | | |
| SF-12 score (vitality) | | | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | VV VV +VV VV | WW WW LWW WW | | |
| Mean ± SD | XX.XX ±XX.XX | XX.XX ±XX.XX | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX<br>Version No.: V1.0 | | 90/120 |
| Medical Research & Biometrics Center, Center for Cardiovascular Diseases | inational | version No.: V1.0 | | 80/129 |
| Control for Carato (aboutar Diboubon | | | | |

| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
|---|---|---|---|---|
| Change in SF-12 score (vitali | ty) relative to before surg | gery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and XX 95% confidence interval | X.XX(XX.XX ,XX.XX) | | | |
| SF-12 score (social functions | ) | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (socia | l functions) relative to be | fore surgery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| interval | | | | |
| | X.XX(XX.XX,XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 40 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery (continued 2)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (emotional conditions) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | XX.XX ±XX.XX | ` ' | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | · · | | |
| Change in SF-12 score (emotional c | · · | · · | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | XX.XX ±XX.XX | • | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | | | |
| Minimum; maximum | XX.XX ;XX.XX | · · | | |
| | 111111111111111111111111111111111111111 | 71717171 ,71717171 | | |
| 95% confidence (XX.) | XX,XX.XX) | (XX.XX, XX.XX) | | |
| The difference and XX.XX(X | (XX.XX, XX.XX | | | |
| 95% confidence | | | | |
| interval | | | | |
| SF-12 score (mental health) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| z Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (mental heal | th) relative to before | re surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | XX.XX ±XX.XX | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence (XX.) | XX,XX.XX) | (XX.XX, XX.XX) | | |
| interval | ,, | () | | |
| · | XX.XX, XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |
| SF-12 score (total physical health so | core) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (total physic | al health score) rela | ative to before surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | XX.XX ±XX.XX | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Medical Research & Biometrics Center, N<br>Center for Cardiovascular Diseases | | Version No.: V1.0 | | 82/129 |

Minimum; maximum XX.XX;XX.XX XX.XX;XX.XX

95% confidence (XX.XX,XX.XX) (XX.XX,XX.XX)
interval

The difference and XX.XX(XX.XX,XX.XX)

95% confidence interval

Notes: 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.

- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 40 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery (continued 3)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (total mental health sco | ore) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (total menta | l health score) relati | ve to before surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence (XX. | .XX ,XX.XX) | (XX.XX,XX.XX) | | |
| interval | | | | |
| The difference and XX.XX( | XX.XX, XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 41 (FAS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Activity level | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Walk easily | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to walk | XXX (XX.X%) | XXX (XX.X%) | | |
| Self-care | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Daily activities (such as work, study, house | work, family or ent | ertainment) | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Pain/discomfort | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Anxiety/depression | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the

intergroup comparison of qualitative indicators;

2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 41 (FAS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 12 weeks after surgery(continue)

| Indicator | Study | group Control gr | oup Statis | tics P value |
|---|---|---|---|---|
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Change in health index rela | tive to before surgery | | | |
| Number of subjects (N miss | s) XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence | (XX.XX, XX.XX) | (XX.XX, XX.XX) | | |
| interval | | | | |
| The difference and $X$ | XX.XX(XX.XX,XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |

Notes:

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 42 (FAS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Activity level | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Walk easily | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to walk | XXX (XX.X%) | XXX (XX.X%) | | |
| Self-care | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Daily activities (such as work, study, house | work, family or ent | ertainment) | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Pain/discomfort | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Anxiety/depression | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the

intergroup comparison of qualitative indicators;

2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 42 (FAS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 24 weeks after surgery(continue)

| Indicator | Study | group | Control grou | ıp Statis | tics P value |
|---|---|---|---|---|---|
| Health index | | | | | |
| Number of subjects (N miss | ) XXX ( | XXX) | XXX (XXX | XXXX | XX X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | XX.XX | $\pm XX.XX$ | | |
| Median | XX.XX | X | X.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX | X;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX | X;XX.XX | | |
| Change in health index relative | to before surgery | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX | (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | XX.XX | $\pm XX.XX$ | | |
| Median | XX.XX | X | X.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX | XXXXX; | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX | X;XX.XX | | |
| 95% confidence (2 | XX.XX ,XX.XX) | (XX.XX | (XX.XX, | | |
| interval | | | | | |
| The difference and XX.X | (XX.XX, XX.XX) | | | | |
| 95% confidence | | | | | |
| interval | | | | | |

Notes:

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

# Table 43 (FAS) Secondary endpoint - Statistical analysis results of subjects' incidence rate of complications requiring re-operation or revision

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Complications requiring re-operation | on or revision | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 44 (PPS) Secondary endpoint - Statistical analysis results of subjects' AE

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total No. | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. Total No.: the number of subjects who occurred AE, if at least once, will be determined as 'Y'
- 2. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 45 (PPS) Secondary endpoint - Statistical analysis results of subjects' revision rate 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Revision 24 weeks after surgery | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 46 (PPS) Secondary endpoint - Statistical analysis results of subjects' re-operation rate 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Re-operation 24 weeks after surgery | 7 | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 47 (PPS) Secondary endpoint - Statistical analysis results of subjects' Harris hip score 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total Harris hip score | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 48 (PPS) Secondary endpoint - Statistical analysis results of subjects' Harris hip score 24 weeks after surgery

| Indicator | | Study group | Control group | Statistics | P value |
|---|---|---|---|---|---|
| Total Harris hip so | core | | | | |
| Number of sumiss) | abjects (N | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | | $XX.XX\pm\!XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | | XX.XX | XX.XX | | |
| Q1; Q3 | | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; m | aximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 49 (FAS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (body function | | | | |
| Number of subjects | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| (N miss) | , , | , | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (bo | ody functions) relative to b | efore surgery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and 95% confidence interval | XX.XX(XX.XX ,XX.X | X) | | |
| SF-12 score (physical cond | ditions) | | | |
| Number of subjects | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| (N miss) | 71111 ( 71111) | 7211 (7211) | 71.71717171 | 11.12 12 12 12 1 |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (pl | nysical conditions) relative | e to before surgery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| 95% confidence interval | X.XX(XX.XX,XX.XX) | | | |
| SF-12 score (body pain) | 373737 / 373737 | 3/3/3/ / 3/3/3/ | 37 37373737 | 37 37373737 |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| · | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 49 (PPS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery (continued 1)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (general health) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (genera | l health) relative to be | efore surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| 95% confidence (X | (XX.XX, XX.XX) | (XX.XX,XX.XX) | | |
| interval | | | | |
| The difference and XX.X 95% confidence interval | X(XX.XX ,XX.XX) | | | |
| SF-12 score (vitality) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (vitality | y) relative to before su | rgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence (Xinterval | (XX.XX, XX.XX) | (XX.XX,XX.XX) | | |
| The difference and XX.X 95% confidence interval | X(XX.XX,XX.XX) | | | |

Version No.: V1.0

96/129

| SF-12 score (social functions) | | | | |
|---|---|---|---|---|
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm \! XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (social to | functions) relative to b | efore surgery | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence (X | X.XX,XX.XX) | (XX.XX,XX.XX) | | |
| interval | | | | |
| The difference and XX.X | X(XX.XX,XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 49 (PPS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery (continued 2)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (emotional con | | <i>⊕</i> r | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | | | |
| Change in SF-12 score (em | * | ŕ | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and XX 95% confidence interval | X.XX(XX.XX,XX.XX) | | | |
| SF-12 score (mental health) | )· | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (me | * | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and XX 95% confidence interval | X.XX(XX.XX ,XX.XX) | | | |
| SF-12 score (total physical | health score) | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Medical Research & Biometrics | Center, National | Version No.: | V1.0 | 98/129 |

Center for Cardiovascular Diseases

| Change in SF-12 score | total phy | sical health score | relative to | before surgery |
|---|---|---|---|---|

| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
|---|---|---|---|---|
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence | (XX.XX, XX.XX) | (XX.XX,XX.XX) | | |

interval

The difference and XX.XX(XX.XX, XX.XX)

95% confidence

interval

Notes:

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 49 (PPS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 12 weeks after surgery (continued 3)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (total mental health se | core) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm\! XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (total ment | tal health score) relat | tive to before surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm \! XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| • | (XXX,XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (XX.XX,XX.XX) | | |
| interval The difference and XX.XX | (XX.XX,XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 50 (PPS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (body functions) | ) | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (body | functions) relative to be | fore surgery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| , | , | , | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and 95% confidence interval | X.XX(XX.XX ,XX.XX) | | | |
| SF-12 score (physical condit | ions) | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (phys | | · · | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX, XX.XX) | | |
| | V VV(VV VV VV VV) | | | |
| 95% confidence interval | X.XX(XX.XX,XX.XX) | | | |
| SF-12 score (body pain) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Medical Research & Biometrics ( | | Version No.: V | 1.0 | 101/129 |
| Tricalcal Research & Diometries | Zenter, rational | v cision ivo V | | 101/129 |

Center for Cardiovascular Diseases

| Change in SF-12 score (body pain) relative to before surgery | | | | |
|---|---|---|---|---|
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and 95% confidence interval | XX.XX(XX.XX ,XX.XX) | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 50 (PPS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery (continued 1)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (general health) | | | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (general hea | alth) relative to befo | re surgery | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| 95% confidence (XX | XX ,XX.XX) | (XX.XX,XX.XX) | | |
| interval | | | | |
| The difference and XX.XX( | XX.XX, XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |
| SF-12 score (vitality) | | | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | $XX.XX \pm \! XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Medical Research & Biometrics Center, Center for Cardiovascular Diseases | National | Version No.: V1.0 | | 102/129 |

| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
|---|---|---|---|---|
| Change in SF-12 score (vitalit | y) relative to before surg | gery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| 95% confidence interval | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| The difference and XX 95% confidence interval | .XX(XX.XX ,XX.XX) | | | |
| SF-12 score (social functions) | | | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | , , | , , | | |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (social | functions) relative to be | fore surgery | | |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX;XX.XX | | |
| 95% confidence | (XX.XX,XX.XX) | (XX.XX,XX.XX) | | |
| interval | | | | |
| | XX(XX,XX,XXX) | | | |
| 95% confidence | | | | |
| interval | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 50 (PPS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery (continued 2)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (emotional conditions) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (emotional | conditions) relative | to before surgery | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| interval | .XX ,XX.XX)<br>XX.XX ,XX.XX) | (XX.XX,XX.XX) | | |
| 95% confidence interval SF-12 score (mental health) | , | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | , , | | |
| Median | XX.XX | XX.XX | | |
| z Q1;Q3 | XX.XX ;XX.XX | | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (mental hea | * | · · | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | XX.XX ±XX.XX | ` ' | | 1 1 1 1 1 1 1 1 1 |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence (XX interval | .XX, XX.XX) | (XX.XX,XX.XX) | | |
| The difference and XX.XX( 95% confidence interval SF-12 score (total physical health s | XX.XX ,XX.XX) | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | XX.XX ±XX.XX | XX.XX ±XX.XX | 211212121 | 11.11111111 |
| Median | XX.XX | XX.XX | | |
| Q1;Q3 | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX ;XX.XX | | |
| Change in SF-12 score (total physic | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | ` ' | 71.71/1/1/1 | 71./1/1/1/1 |
| Median | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Q1;Q3 | | XX.XX ;XX.XX | | |
| Medical Research & Biometrics Center, | XX.XX ;XX.XX National | Version No.: V1.0 | | 104/129 |
| Center for Cardiovascular Diseases | | | | |

Minimum; maximum XX.XX;XX.XX XX.XX;XX.XX

95% confidence (XX.XX,XX.XX) (XX.XX,XX.XX)
interval

The difference and XX.XX(XX.XX,XX.XX)
95% confidence
interval

Notes: 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.

- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 50 (PPS) Secondary endpoint - Statistical analysis results of subjects' SF-12v2 questionnaire 24 weeks after surgery (continued 3)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| SF-12 score (total mental health score) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Change in SF-12 score (total mental health score) relative to before surgery | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX\pm\!XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX ;XX.XX | XX.XX;XX.XX | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX ;XX.XX | | |
| 95% confidence (XX. | .XX,XX.XX) | (XX.XX, XX.XX) | | |
| interval | | | | |
| ` | XX.XX, XX.XX) | | | |
| 95% confidence | | | | |
| interval | | | | |

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 51 (PPS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Activity level | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Walk easily | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to walk | XXX (XX.X%) | XXX (XX.X%) | | |
| Self-care | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Daily activities (such as work, study, housework, family or entertainment) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Pain/discomfort | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Anxiety/depression | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the
intergroup comparison of qualitative indicators;

2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 51 (PPS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 12 weeks after surgery(continue)

| Indicator | Study | group | Control grou | ıp Statis | stics P v | alue |
|---|---|---|---|---|---|---|
| Health index | | | | | | |
| Number of subjects (N mis | s) XXX ( | XXX) | XXX (XXX | XXX | XXX X.X | XXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | XX.XX | $X \pm XX.XX$ | | | |
| Median | XX.XX | X | X.XX | | | |
| Q1; Q3 | XX.XX;XX.XX | XX.X | X ;XX.XX | | | |
| Minimum; maximum | XX.XX;XX.XX | XX.X | X ;XX.XX | | | |
| Change in health index relative | to before surgery | | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX | X (XXX) | X.XXXX | X.XXXX | |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | XX.XX | $X \pm XX.XX$ | | | |
| Median | XX.XX | X | X.XX | | | |
| Q1; Q3 | XX.XX;XX.XX | XX.X | X ;XX.XX | | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.X | X ;XX.XX | | | |
| 95% confidence ( | (XX.XX, XX.XX) | (XX.XX | X,XX.XX) | | | |
| interval | | | | | | |
| The difference and XX. | XX(XX.XX, XX.XX) | | | | | |
| 95% confidence | | | | | | |
| interval | | | | | | |

#### Notes:

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 52 (PPS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Activity level | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Walk easily | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in walking | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to walk | XXX (XX.X%) | XXX (XX.X%) | | |
| Self-care | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in washing or dressing independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to wash or dress independently | XXX (XX.X%) | XXX (XX.X%) | | |
| Daily activities (such as work, study, house | work, family or ent | ertainment) | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Easy to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Slightly difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Very difficult in performing daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Completely unable to perform daily activities | XXX (XX.X%) | XXX (XX.X%) | | |
| Pain/discomfort | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe pain/discomfort | XXX (XX.X%) | XXX (XX.X%) | | |
| Anxiety/depression | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Moderate anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |
| Very severe anxiety/depression | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the

intergroup comparison of qualitative indicators;

2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);;

Table 52 (PPS) Secondary endpoint - Statistical analysis results of subjects' EQ-5D questionnaire 24 weeks after surgery(continue)

| Indicator | Study | group | Control gro | up Stat | istics | P value |
|---|---|---|---|---|---|---|
| Health index | | | | | | |
| Number of subjects (N mis | ss) XXX ( | XXX) | XXX (XXX | X) X.X | XXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | XX.XX | $X \pm XX.XX$ | | | |
| Median | XX.XX | X | X.XX | | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX | X;XX.XX | | | |
| Minimum; maximum | XX.XX;XX.XX | XX.XX | X ;XX.XX; | | | |
| Change in health index relative | e to before surgery | | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX | (XXX) | X.XXXX | X.2 | XXXX |
| $Mean \pm SD$ | $XX.XX\pm\!XX.XX$ | XX.XX | $X \pm XX.XX$ | | | |
| Median | XX.XX | X | X.XX | | | |
| Q1; Q3 | XX.XX;XX.XX | XX.XX | X ;XX.XX; | | | |
| Minimum; maximum | XX.XX ;XX.XX | XX.XX | X;XX.XX | | | |
| 95% confidence | (XX.XX,XX.XX) | (XX.XX | (XX.XX, | | | |
| interval | | | | | | |
| The difference and XX. | XX(XX.XX, XX.XX) | | | | | |
| 95% confidence | | | | | | |
| interval | | | | | | |

Notes:

- 1. Group t-test or Wilcoxon rank-sum test is used to analyze the intergroup comparison of quantitative indicators.
- 2. In quantitative indicators, Q1: 25th quantile, Q3: 75th percentile.
- 3. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 53 (PPS) Secondary endpoint - Statistical analysis results of subjects' incidence rate of complications requiring re-operation or revision

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Complications requiring re-operation | on or revision | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 54 Statistical analysis results of subjects' AE evaluation 1 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether there are adverse events or | complications in the | subjects after the last | follow-up | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 55 Statistical analysis results of subjects' medication records 1 week after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new drugs are added to the concomitant medication or whether the original concomitant | | | | |
| medication is changed | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 56 Statistical analysis results of subjects' combination therapy 1 week after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new types of combination the | rapy are added | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 57 Statistical analysis results of subjects' fractures 1 week after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Wound healing - healing grade | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A | XXX (XX.X%) | XXX (XX.X%) | | |
| В | XXX (XX.X%) | XXX (XX.X%) | | |
| C | XXX (XX.X%) | XXX (XX.X%) | | |
| Wound healing - incision category | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I | XXX (XX.X%) | XXX (XX.X%) | | |
| Class II | XXX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Focal tenderness | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe | XXX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Lengthwise percussion | pain | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe | XXX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Abnormal activity | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Evaluate postoperative weight-bearing | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No weight-bearing | XXX (XX.X%) | XXX (XX.X%) | | |
| Lower degree of weight-bearing (support with two crutches) | XXX (XX.X%) | XXX (XX.X%) | | |
| Higher degree of weight-bearing (support with one crutch) | XXX (XX.X%) | XXX (XX.X%) | | |
| Fully weight-bearing (support without crutch) | XXX (XX.X%) | XXX (XX.X%) | | |
| After the investigational device is impl stability of the fracture site | anted, whether exte | rnal fixation is requ | ired to enhanc | e the |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 58 Statistical analysis results of subjects' x-ray examination at the fracture site 1 week after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Reduction | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Stable | XXX (XX.X%) | XXX (XX.X%) | | |
| Loss of reduction | XXX (XX.X%) | XXX (XX.X%) | | |
| Is the re-operation required | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Implant | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of intramedullary nail | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of | XXX (XX.X%) | XXX (XX.X%) | | |
| intramedullary nail | | | | |
| Fracture line | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Clear | XXX (XX.X%) | XXX (XX.X%) | | |
| Vague | XXX (XX.X%) | XXX (XX.X%) | | |
| Disappeared | XXX (XX.X%) | XXX (XX.X%) | | |
| Callus | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Intermittent | XXX (XX.X%) | XXX (XX.X%) | | |
| Continuous | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 59 Statistical analysis results of subjects' AE evaluation 6 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether there are adverse events or o | complications in the | subjects after the last | follow-up | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 60 Statistical analysis results of subjects' medication records 6 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new drugs are added to the c medication is changed | oncomitant medicati | on or whether the or | riginal concon | nitant |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 61 Statistical analysis results of subjects' combination therapy 6 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new types of combination the | nerapy are added | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 62 Statistical analysis results of subjects' fractures 6 weeks after surgery

| Indicator S | Study group | Control group | Statistics | - 1 |
|---|---|---|---|---|
| | | Control group | Statistics | P value |
| Wound healing - healing grade | | | | |
| Number of subjects (N miss) | XX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A X | XX (XX.X%) | XXX (XX.X%) | | |
| B | XX (XX.X%) | XXX (XX.X%) | | |
| C | XX (XX.X%) | XXX (XX.X%) | | |
| Wound healing - incision category | | | | |
| Number of subjects (N miss) | XX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I X | XX (XX.X%) | XXX (XX.X%) | | |
| Class II X | XX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Focal tenderness | | | | |
| Number of subjects (N miss) | XX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA X | XX (XX.X%) | XXX (XX.X%) | | |
| Mild | XX (XX.X%) | XXX (XX.X%) | | |
| Severe XX | XX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Lengthwise percussion pain | | | | |
| Number of subjects (N miss) X | XX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA X | XX (XX.X%) | XXX (XX.X%) | | |
| Mild | XX (XX.X%) | XXX (XX.X%) | | |
| Severe XX | XX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Abnormal activity | | | | |
| Number of subjects (N miss) | XX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes X | XX (XX.X%) | XXX (XX.X%) | | |
| No X | XX (XX.X%) | XXX (XX.X%) | | |
| Evaluate postoperative weight-bearing | | | | |
| Number of subjects (N miss) X | XX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No weight-bearing XX | XX (XX.X%) | XXX (XX.X%) | | |
| Lower degree of weight-bearing (support with two crutches) | XX (XX.X%) | XXX (XX.X%) | | |
| Higher degree of weight-bearing (support with one crutch) | XX (XX.X%) | XXX (XX.X%) | | |
| Fully weight-bearing (support without crutch) | XX (XX.X%) | XXX (XX.X%) | | |
| After the investigational device is implanted stability of the fracture site | l, whether extern | nal fixation is requir | ed to enhance | the |
| - | XX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| • | XX (XX.X%) | XXX (XX.X%) | | |
| | XX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 63 Statistical analysis results of subjects' X-ray examination at the fracture site 6 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Reduction | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Stable | XXX (XX.X%) | XXX (XX.X%) | | |
| Loss of reduction | XXX (XX.X%) | XXX (XX.X%) | | |
| Is the re-operation required | , , | , , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Implant | , | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of intramedullary nail | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of intramedullary nail | XXX (XX.X%) | XXX (XX.X%) | | |
| Fracture line | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Clear | XXX (XX.X%) | XXX (XX.X%) | | |
| Vague | XXX (XX.X%) | XXX (XX.X%) | | |
| Disappeared | XXX (XX.X%) | XXX (XX.X%) | | |
| Callus | , , | , , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Intermittent | XXX (XX.X%) | XXX (XX.X%) | | |
| Continuous | XXX (XX.X%) | XXX (XX.X%) | | |
| The frontal/lateral X-ray examination | shows the continuou | us callus passing acr | oss the fractur | e line |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Determine the fracture union condition | ` ' | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No union | XXX (XX.X%) | XXX (XX.X%) | | |
| Union | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 64 Statistical analysis results of subjects' AE evaluation 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether there are adverse events or co | omplications in the st | abjects after the last | follow-up | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 65 Statistical analysis results of subjects' medication records 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new drugs are added to the concomitant medication or whether the original concomitant | | | | |
| medication is changed | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 66 Statistical analysis results of subjects' combination therapy 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new types of combination the | erapy are added | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 67 Statistical analysis results of subjects' fractures 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Wound healing - healing grade | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A | XXX (XX.X%) | XXX (XX.X%) | | |
| В | XXX (XX.X%) | XXX (XX.X%) | | |
| С | XXX (XX.X%) | XXX (XX.X%) | | |
| Wound healing - incision category | ` , | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I | XXX (XX.X%) | XXX (XX.X%) | | |
| Class II | XXX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Focal tenderness | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe | XXX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Lengthwise percussion | pain | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Mild | XXX (XX.X%) | XXX (XX.X%) | | |
| Severe | XXX (XX.X%) | XXX (XX.X%) | | |
| Physical sign - Abnormal activity | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Evaluate postoperative weight-bearing | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No weight-bearing | XXX (XX.X%) | XXX (XX.X%) | | |
| Lower degree of weight-bearing (support with two crutches) | XXX (XX.X%) | XXX (XX.X%) | | |
| Higher degree of weight-bearing (support with one crutch) | XXX (XX.X%) | XXX (XX.X%) | | |
| Fully weight-bearing (support without crutch) | XXX (XX.X%) | XXX (XX.X%) | | |
| After the investigational device is impl<br>stability of the fracture site | anted, whether exte | rnal fixation is requi | red to enhance | e the |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | _ | _ |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 68 Statistical analysis results of subjects' X-ray examination at the fracture site 12 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Reduction | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Stable | XXX (XX.X%) | XXX (XX.X%) | | |
| Loss of reduction | XXX (XX.X%) | XXX (XX.X%) | | |
| Is the re-operation required | , | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Implant | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of intramedullary nail | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of intramedullary | XXX (XX.X%) | XXX (XX.X%) | | |
| nail | | | | |
| Fracture line | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Clear | XXX (XX.X%) | XXX (XX.X%) | | |
| Vague | XXX (XX.X%) | XXX (XX.X%) | | |
| Disappeared | XXX (XX.X%) | XXX (XX.X%) | | |
| Callus | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Intermittent | XXX (XX.X%) | XXX (XX.X%) | | |
| Continuous | XXX (XX.X%) | XXX (XX.X%) | | |
| The frontal/lateral X-ray examination | shows the continuo | us callus passing acr | oss the fractur | e line |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Determine the fracture union condition | n | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No union | XXX (XX.X%) | XXX (XX.X%) | | |
| Union | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 69 Statistical analysis results of subjects' AE evaluation 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether there are adverse events or co | omplications in the s | ubjects after the last | follow-up | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX<br>(XX.X%) | XXX (XX.X%) | | |
| No | XXX<br>(XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 70 Statistical analysis results of subjects' medication records 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new drugs are added to the concomitant medication or whether the original concomitant medication is changed | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 71 Statistical analysis results of subjects' combination therapy 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Whether new types of combination the | erapy are added | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 72 Statistical analysis results of subjects' fractures 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Wound healing - healing grade | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| В | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| С | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Wound healing - incision category | | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Class II | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Physical sign - Focal tenderness | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Mild | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Severe | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Physical sign - Lengthwise percussion | n pain | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Mild | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Severe | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Physical sign - Abnormal activity | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| No | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Evaluate postoperative weight-bearing | g | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No weight-bearing | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Lower degree of weight-bearing (support with two crutches) | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Higher degree of weight-<br>bearing (support with one<br>crutch) | XXX (XX.X%) | XXX<br>(XX.X%) | | |
| Fully weight-bearing (support without crutch) | XXX (XX.X%) | XXX<br>(XX.X%) | | |

After the investigational device is implanted, whether external fixation is required to enhance the

| stability of the fracture site | | | | |
|--------------------------------|-------------|-----------|--------|--------|
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX | | |
| | | (XX.X%) | | |
| No | XXX (XX.X%) | XXX | | |
| | | (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 73 Statistical analysis results of subjects' x-ray examination at the fracture site 24 weeks after surgery

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Reduction | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Stable | XXX (XX.X%) | XXX (XX.X%) | | |
| Loss of reduction | XXX (XX.X%) | XXX (XX.X%) | | |
| Is the re-operation required | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Implant | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Rupture of intramedullary nail | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of screw/bolt | XXX (XX.X%) | XXX (XX.X%) | | |
| Displacement of intramedullary nail | XXX (XX.X%) | XXX (XX.X%) | | |
| Fracture line | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Clear | XXX (XX.X%) | XXX (XX.X%) | 71.71717171 | 21.212121 |
| Vague | XXX (XX.X%) | XXX (XX.X%) | | |
| Disappeared | XXX (XX.X%) | XXX (XX.X%) | | |
| Callus | 7222 (722.7170) | 71711 (7171.7170) | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Intermittent | XXX (XX.X%) | XXX (XX.X%) | | |
| Continuous | XXX (XX.X%) | XXX (XX.X%) | | |
| The frontal/lateral X-ray examination | , , , | , | oss the fracture | line |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Determine the fracture union condition | ` ' | , | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No union | XXX (XX.X%) | XXX (XX.X%) | | |
| Union | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 74 Statistical analysis results of outcomes of subjects' complete blood count before and after surgery (before surgery → immediately after surgery)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| White blood cell (WBC) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal $\rightarrow$ Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| NE | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal $\rightarrow$ Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Red blood cell (RBC) | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| HGB | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal $\rightarrow$ Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| Platelet | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal $\rightarrow$ Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal → Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 74 Statistical analysis results of outcomes of subjects' complete blood count before and after surgery (before surgery → immediately after surgery) (continued)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| INR | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| APTT | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 75 List of subjects with abnormal complete blood count with clinical significance after surgery changed from normal indicators before surgery (before surgery → immediately after surgery)

| Indicator | Site No. | Random<br>No. | Group | Age | Gender | Before<br>surgery | Immediately<br>after surgery |
|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX |

Table 76 Statistical analysis results of outcomes of subjects' blood biochemical test before and after surgery (before surgery → immediately after surgery)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| AST | Study group | Control group | Statistics | r value |
| Number of subjects (N miss) | XXX ( XXX) | XXX ( XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical | , , | • | 71.71.71.71.71 | 71.71.71.71 |
| significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| ALT | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| ALB | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| CHOL | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal → Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| TRIG | () | () | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal → Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 76 Statistical analysis results of outcomes of subjects' blood biochemical test before and after surgery (before surgery → immediately after surgery) (continued 1)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| CREA | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| BUN | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| UREA | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| UA | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| LDL-C | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 76 Statistical analysis results of outcomes of subjects' blood biochemical test before and after surgery (before surgery → immediately after surgery) (continued 2)

| Indicator | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| HDL-C | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| GLU | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| $Normal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| CRP | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal $\rightarrow$ Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Abnormal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Hypersensitive CRP | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal → Abnormal (with clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Abnormal (without clinical significance) | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal → Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| $Abnormal \rightarrow Normal$ | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal → Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 77 List of subjects with abnormal blood biochemical test indicators with clinical significance after surgery changed from normal indicators before surgery (before surgery → immediately after surgery)

| Indicator | Site No. | Random<br>No. | Group | Age | Gender | Before<br>surgery | Immediately after surgery |
|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX |

 Table 78
 List of concomitant medication of subjects

| Site<br>No. | Random<br>No. | Group | Age | Gender | Drug<br>name | Indication<br>or reason<br>for<br>medication | For<br>treating<br>AE | Single<br>dose | Unit | Frequency of administration per day | Route of administration | Start date of administration | End date of administration | Still use after<br>completion of<br>the trial |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | | | | ••••• | | | | | | | |
| ••••• | | | • | | | ••••• | • | ••••• | | | | | | |
Table 79 Specific description on subjects with AEs

| Site<br>No. | Random<br>No. | Group | Age | Gender | Name<br>of AE<br>(SOC<br>code) | Name<br>of AE<br>(PT<br>code) | Time of<br>postoperative<br>occurrence<br>(day) | Remission<br>time (day) | Severity | Measures<br>taken | Outcome | Correlation with the surgery | Correlation<br>with the<br>investigational<br>device | Withdrawal<br>from the<br>trial due to<br>AEs | Whether<br>it is<br>UADE | Whether<br>it is<br>device<br>failure | Whether<br>it is<br>SAE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

1. Time of postoperative occurrence (day) = Date of occurrence of AE - Date of surgery; Remission time (day) = End date of AE - Date of occurrence of AE.

Table 80 Summary of AEs

| Adverse event | S | tudy group | Contr | rol group |
|---|---|---|---|---|
| | Number of events | Number of subjects (N=XXX) | Number of events | Number of<br>subjects<br>(N=XXX) |
| Name of AE (SOC code) | XXX | XXX(XX.XX% <sup>#</sup> ) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | | | | |
| Name of AE (SOC code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | | | | |

- 1. #: Percentage of AEs = Number of subjects suffering from AEs/Total number of subjects in the study group or the control group;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

**Table 80 Summary of AEs (continued 1)** 

| Adverse event | Study group | Control group | Statistics | P value |
|-----------------------|-------------|---------------|------------|---------|
| Total number of AEs | | | | |
| Number of subjects (N | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| miss) | | | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

Event rate difference (study group-control group) and 95%CI XX.X [XX.X; XX.X]

Notes:

- 1. The total number of AEs refers to the number of subjects suffering from AEs, and the AEs occur in the subject at least one time, which is considered as "Yes".
- 2. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 3. The difference of event rate and 95% confidence interval were analyzed by Wald test with continuous correction;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 81 Specific description on subjects with investigational device-related AEs

| Site No. | Random<br>No. | Group | Age | Gender | Name of<br>AE<br>(SOC<br>code) | Name of<br>AE (PT<br>code) | Time of postoperative occurrence (day) | Remission<br>time (day) | Severity | Measures<br>taken | Outcome | Correlation<br>with the<br>surgery | Correlation<br>with the<br>investigational<br>device | Withdrawal<br>from the<br>trial due to<br>AEs | Whether<br>it is<br>UADE | Whether<br>it is<br>device<br>failure | Whether |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes:

1. Time of postoperative occurrence (day) = Date of occurrence of AE - Date of surgery; Remission time (day) = End date of AE - Date of occurrence of AE

Table 82 Summary of investigational device-related AEs

| Investigational device-<br>related AE | Str | udy group | Control group | |
|---|---|---|---|---|
| | Number of events | Number of subjects (N=XXX) | Number of events | Number of subjects (N=XXX) |
| Name of AE (SOC code) | XXX | XXX(XX.XX% <sup>#</sup> ) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | | | | |
| Name of AE (SOC code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of AE (PT code) | | | | |

- 1. #: Percentage of investigational device-related AEs = Number of subjects suffering from investigational device-related AEs/Total number of subjects in the study group or the control group;
- 2: Investigational device-related AEs refer to those "definitely related", "probably related" and "possibly related" with the investigational device;
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 82 Summary of investigational device-related AEs (continued)

| Investigational device-related AE | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total number of investigational device- | elated AEs | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Event rate difference (study group-contro | l group) and 95%CI | XX.X [XX.X; | XX.X] | |

- 1. The total number of investigational device-related AEs refers to the number of subjects suffering from investigational device-related AEs and the investigational device-related AEs occur in the subject at least one time, which is considered as "Yes".
- 2: Investigational device-related AEs refer to those "definitely related", "probably related" and "possibly related" with the investigational device;
- 3. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 4. The difference of event rate and 95% confidence interval were analyzed by Wald test with continuous correction;
- 5. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

# Table 83 Summary of AEs (Number of events per subject)

Study group  $(N=XXX^{\#1})$  control group  $(N=XXX^{\#1})$ P Indicator Total number of adverse events XXX #2( XX.X <sup>3</sup>) XXX #2 ( XX.X <sup>#3</sup>) X.XXXX Event difference (study group-control group) and 95%C XX.X [XX.X; XX.X] Total number of device related adverse events  $XXX^{\#2}(XX.X^{3})$   $XXX^{\#2}(XX.X^{\#3})$ X.XXXX Event rate difference (study group-control group) and 95%CI XX.X [XX.X; XX.X] Total number of surgery related adverse events  $XXX^{\#2}(XX.X^3) XXX^{\#2}(XX.X^{\#3})$ X.XXXX Event rate difference (study group-control group) and 95%CI XX.X [XX.X; XX.X] Notes: 1. Devices related adverse events are the adverse events that are "probably related" or "possible

related" or "definitely related" to the study devices;

- 3.#1: Total number of subjects; #2: Total number of events;
  - #3: Total number of events/total number of patients: the average number of events per subject;
- 4. Group t-test is used to analyze Event rate difference (study group-control group) and 95%CI
- 5. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

<sup>2.</sup> Surgery related adverse events are the adverse events that are "probably related" or "possible related" or "definitely related" to surgery;

Table 84 Statistical analysis results of the severity and the device related AEs (According subject)

| Indicator | Study group control gr | roup statistic | P | |
|---|---|---|---|---|
| Severity | | | | |
| NO. (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| mild | XXX (XX.X%) | XXX (XX.X% | (b) | |
| moderate | XXX (XX.X%) | XXX (XX.Xº | %) | |
| severe | XXX (XX.X%) | XXX (XX.X | (%) | |
| Device related | | | | |
| NO. (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Not related | XXX (XX.X | %) XXX (X | (X.X%) | |
| Unlikely related | XXX (XX.X | %) XXX (X | (X.X%) | |
| Possible related | XXX (XX.X% | ) XXX (XX | X.X%) | |
| probably related | XXX (XX.X%) | ) XXX (XX | (.X%) | |
| definitely related | XXX (XX.Xº | %) XXX (X | (X.X%) | |
| Surgery related | | | | |
| NO. (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Not related | XXX (XX.X% | (6) XXX (X | X.X%) | |
| Unlikely related | XXX (XX.X | %) XXX (X | (X.X%) | |
| possible related | XXX (XX.X% | ) XXX (XX | (XX%) | |
| probably related | XXX (XX.X%) | ) XXX (XX | (.X%) | |
| definitely related | XXX (XX.X | X%) XXX ( | XX.X%) | |

Notes: 1. If more than one adverse event occurred in a subject, the analysis was performed with the highest severity or correlation;

<sup>2.</sup> The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;

<sup>3.</sup> Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 85 Statistical analysis results of the severity and the device related AEs (Number of events per subject)

| Indicator<br>(N=XXX#1) | Study group (N=XXX#1) | control group(N | I=XXX#1) total |
|---|---|---|---|
| Severity | | | |
| mild | XXX#2 (XX.X%#3) | XXX (XX.X%) | XXX (XX.X%) |
| moderate | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| severe | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Device related | | | |
| Not related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Unlikely related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Possible related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| probably related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| definitely related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Surgery related | | | |
| Not related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Unlikely related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| possible related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| probably related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| definitely related | XXX (XX.X% | S) XXX (XX.X% | (X, X, X |

Notes: 1.#1: Total number of subjects; #2: Total number of events;

<sup>2.#3:</sup> Total number of events/total number of subjects: the average number of events per subject;

<sup>3.</sup> Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II)

Table 86 Specific description on subjects with SAEs

| Site<br>No. | Random<br>No. | Group | Age | Gender | Name<br>of<br>SAE<br>(SOC<br>code) | Name<br>of<br>SAE<br>(PT<br>code) | Time of postoperative occurrence (day) | Remission<br>time (day) | Severity | Outcome | Correlation with the surgery | Correlation<br>with the<br>investigational<br>device | SAE<br>condition |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes: 1. Time of postoperative occurrence (day) = Date of occurrence of SAE - Date of surgery; Remission time (day) = End date of SAE - Date of occurrence of SAE.

**Table 87 Summary of SAEs** 

| SAE | Stı | ıdy group | Cont | rol group |
|---|---|---|---|---|
| | Number of events | Number of subjects (N=XXX) | Number of events | Number of subjects (N=XXX) |
| Name of SAE (SOC code) | XXX | $XXX(XX.XX\%^{\#})$ | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | | | | |
| Name of SAE (SOC code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | | | | |

- 1. #: Percentage of SAEs = Number of subjects suffering from SAEs/Total number of subjects in the study group or the control group;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

# **Table 87 Summary of SAEs (continued)**

| SAE | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total number of SAEs | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

Event rate difference (investigation group-control group) and 95%CI XX.X [XX.X; XX.X]

Notes:

- 1. The total number of SAEs refers to the number of subjects suffering from SAEs and the SAEs occur in the subject at least one time, which is considered as "Yes".
- 2. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 3. The difference of event rate and 95% confidence interval were analyzed by Wald test with continuous correction;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 88 Specific description on subjects with investigational device-related SAEs

| Site<br>No. | Random<br>No. | Group | Age | Gender | Name<br>of<br>SAE<br>(SOC<br>code) | Name<br>of<br>SAE<br>(PT<br>code) | Time of postoperative occurrence (day) | Remission<br>time (day) | Severity | Outcome | Correlation with the surgery | Correlation<br>with the<br>investigational<br>device | SAE<br>condition |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes: 1. Time of postoperative occurrence (day) = Date of occurrence of SAE - Date of surgery; Remission time (day) = End date of SAE - Date of occurrence of SAE.

Table 89 Summary of investigational device-related SAEs

| | S1 | udy group | Control group | |
|---|---|---|---|---|
| Investigational device-related SAE | Number of events | Number of subjects (N=XXX) | Number of events | Number of<br>subjects<br>(N=XXX) |
| Name of SAE (SOC code) | XXX | XXX(XX.XX% <sup>#</sup> ) | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | | | | |
| Name of SAE (SOC code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of SAE (PT code) | | | | |

- 1. #: Percentage of investigational device-related SAEs = Number of subjects suffering from investigational device-related SAEs/Total number of subjects in the study group or the control group;
- 2: Investigational device-related SAEs refer to those "definitely related", "probably related" and "possibly related" with the investigational device;
- 3. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 89 Summary of investigational device-related SAEs (continued)

| Investigational related SAE | device- | Study group | Control group | Statistics | P value |
|---|---|---|---|---|---|
| Total number of investigational devrelated SAEs | rice- | | | | |
| Number of subjects | s (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | | XXX (XX.X%) | XXX (XX.X%) | | |
| No | | XXX (XX.X%) | XXX (XX.X%) | | |
| Event rate difference | e (investiga | XX.X [XX.X; X | XX.X] | | |

- 1. The total number of investigational device-related SAEs refers to the number of subjects suffering from investigational device-related SAEs and the investigational device-related SAEs occur in the subject at least one time, which is considered as "Yes".
- 2: Investigational device-related SAEs refer to those "definitely related", "probably related" and "possibly related" with the investigational device;
- 3. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 4. The difference of event rate and 95% confidence interval were analyzed by Wald test with continuous correction;
- 5. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

## Table 90 Summary of SAEs (Number of events per subject)

Study group  $(N=XXX^{\#1})$  control group  $(N=XXX^{\#1})$ P Indicator Total number of adverse events XXX #2( XX.X <sup>3</sup>) XXX #2 ( XX.X <sup>#3</sup>) X.XXXX Event difference (study group-control group) and 95%C XX.X [XX.X; XX.X] Total number of device related adverse events X.XXXX Event rate difference (study group-control group) and 95%CI XX.X [XX.X; XX.X] Total number of surgery related adverse events X.XXXX Event rate difference (study group-control group) and 95%CI XX.X [XX.X; XX.X] ..... Notes: 1. Devices related adverse events are the adverse events that are "probably related" or "possible

- related" or "definitely related" to the study devices;
- 2. Surgery related adverse events are the adverse events that are "probably related" or "possible related" or "definitely related" to surgery;
- 3.#1: Total number of subjects; #2: Total number of events;
  - #3: Total number of events/total number of patients: the average number of events per subject;
- 4. Group t-test is used to analyze Event rate difference (study group-control group) and 95%CI
- 5. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 91 Statistical analysis results of the severity and the device related SAEs (According subject)

| Indicator | Study group control gr | oup statistic | P | |
|---|---|---|---|---|
| Severity | | | | |
| NO. (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| mild | XXX (XX.X%) | XXX (XX.X% | <b>b</b> ) | |
| moderate | XXX (XX.X%) | XXX (XX.Xº | %) | |
| severe | XXX (XX.X%) | XXX (XX.X | (%) | |
| Device related | | • | | |
| NO. (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Not related | XXX (XX.X <sup>c</sup> | %) XXX (X | (X.X%) | |
| Unlikely related | XXX (XX.X <sup>c</sup> | %) XXX (X | (X.X%) | |
| Possible related | XXX (XX.X%) | ) XXX (XX | (XX%) | |
| probably related | XXX (XX.X%) | XXX (XX | (.X%) | |
| definitely related | XXX (XX.X% | (6) XXX (X | (X.X%) | |
| Surgery related | | | | |
| NO. (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Not related | XXX (XX.X% | ) XXX (XX | X.X%) | |
| Unlikely related | XXX (XX.X <sup>c</sup> | %) XXX (X | (X.X%) | |
| possible related | XXX (XX.X%) | ) XXX (XX | (.X%) | |
| probably related | XXX (XX.X%) | XXX (XX | (.X%) | |
| definitely related | XXX (XX.X | (%) XXX (? | XX.X%) | |

Notes: 1. If more than one adverse event occurred in a subject, the analysis was performed with the highest severity or correlation;

<sup>2.</sup> The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;

<sup>3.</sup> Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

Table 92 Statistical analysis results of the severity and the device related SAEs (Number of events per subject)

Study group (N=XXX#1) control group (N=XXX#1) Indicator total (N=XXX#1)Severity mild XXX#2 (XX.X%#3) XXX (XX.X%) XXX (XX.X%) moderate XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) severe XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) Device related Not related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) Unlikely related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) Possible related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) probably related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) definitely related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) Surgery related Not related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) Unlikely related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) possible related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) probably related XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) definitely related XXX (XX.X%) XXX (XX.X%)

Notes: 1.#1: Total number of subjects; #2: Total number of events;

<sup>2.#3:</sup> Total number of events/total number of subjects: the average number of events per subject;

<sup>3.</sup> Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II)

 Table 93
 Specific description on subjects with UADEs

| Site No. | Random<br>No. | Group | Age | Gender | Name<br>of AE<br>(SOC<br>code) | Name<br>of AE<br>(PT<br>code) | Time of postoperative occurrence (day) | Remission<br>time (day) | Severity | Measures<br>taken | Outcome | Correlation with the surgery | Correlation<br>with the<br>investigational<br>device | Withdrawal<br>from the<br>trial due to<br>AEs | Whether<br>it is<br>device<br>failure | Whether it is SAE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

1. Time of postoperative occurrence (day) = Date of occurrence of AE - Date of surgery; Remission time (day) = End date of AE - Date of occurrence of AE.

**Table 94 Summary of UADEs** 

| UADE | S | tudy group | Со | Control group |
|---|---|---|---|---|
| | Number of events | Number of subjects (N=XXX) | Number of events | Number of subjects (N=XXX) |
| Name of adverse reaction (SOC code) | XXX | XXX(XX.XX% <sup>#</sup> ) | XXX | XXX(XX.XX%) |
| Name of adverse reaction (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of adverse reaction (PT code) | | | | |
| Name of adverse reaction (SOC code) | XXX | $XXX(XX.XX\%^{\#})$ | XXX | XXX(XX.XX%) |
| Name of adverse reaction (PT code) | XXX | XXX(XX.XX%) | XXX | XXX(XX.XX%) |
| Name of adverse reaction (PT code) | | | | |

- 1. #: Percentage of adverse reactions = Number of subjects suffering from adverse reactions/Total number of subjects in the study group or the control group;
- 2. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II);

**Table 94 Summary of UADEs (continued)** 

| UADE | Study group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total number of UADEs | | | | |
| Number of subjects (N miss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

Event rate difference (investigation group-control group) and 95%CI XX.X [XX.X; XX.X]

Notes:

- 1. The total number of UADEs refers to the number of subjects suffering from UADE, and the UADE occur in the subject at least one time, which is considered as "Yes".
- 2. The likelihood ratio Chi-square test or Fisher's exact probability test is used to analyze the intergroup comparison of qualitative indicators;
- 3. The difference of event rate and 95% confidence interval were analyzed by Wald test with continuous correction;
- 4. Investigational device: Trochanteric Fixation Nail Advanced (TFNA); control device: Proximal Femoral Nail Antirotation (PFNA-II)